CLINICAL TRIAL: NCT00083889
Title: A Phase 3, Randomized Study Of SU011248 Versus Interferon-Alfa As First-Line Systemic Therapy For Patients With Metastatic Renal Cell Carcinoma
Brief Title: SU011248 Versus Interferon-Alfa As First-Line Systemic Therapy For Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181034; NCT00098657 (obsolete NCT alias)
Record Dates: First submitted 2004-06-03; First posted 2004-06-04 (Estimated); Results first posted 2009-12-10 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interferon-alpha; Interferon alpha-2; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Interferon-alfa
- 1 (Experimental)
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: Interferon-alfa — 3 MIU first week, 6 MIU second week, and 9 MIU thereafter three times a week (non-consecutive days) until progression or unacceptable toxicity
  Other Names: Roferon
  Arms: 2
Drug: SU011248 — 50 mg orally daily for 4 weeks and 2 weeks off treatment until progression or unacceptable toxicity
  Other Names: Sunitinib, SUTENT
  Arms: 1

SUMMARY:
The purpose of this study is to test whether SU011248 has activity and is safe compared to interferon-alfa as first-line therapy in patients with metastatic renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma of clear cell histology with metastases
* Evidence of measurable disease by radiographic technique
* Eastern Cooperative Oncology Group [ECOG] performance status of 0 or 1

Exclusion Criteria:

* Prior systemic (including adjuvant or neoadjuvant) therapy of any kind for RCC
* History of or known brain metastases
* Serious acute or chronic illness or recent history of significant cardiac abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2004-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (98):
- United States (44):
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detoit, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Australia (7):
  - Pfizer Investigational Site, Lismore, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, South Brisbane, Queensland
  - Pfizer Investigational Site, Woodville South, South Australia
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
  - Pfizer Investigational Site, Victoria
- Brazil (2):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
- Canada (9):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- France (6):
  - Pfizer Investigational Site, Paris, Cedex 15
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Ulm
- Italy (4):
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Roma
- Poland (8):
  - Pfizer Investigational Site, Moczowego, Warszawa
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Russia (5):
  - Pfizer Investigational Site, Obninsk, Kaluga Oblast
  - Pfizer Investigational Site, Chelyabinsk
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Tomsk
- Spain (4):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Seville, SEVILLA
- United Kingdom (5):
  - Pfizer Investigational Site, Whitchurch, Cardiff
  - Pfizer Investigational Site, Manchester, Lancashire
  - Pfizer Investigational Site, Northwood, Middlesex
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Sutton Surrey

REFERENCES:
- [Derived] Rini BI, Hutson TE, Figlin RA, Lechuga MJ, Valota O, Serfass L, Rosbrook B, Motzer RJ. Sunitinib in Patients With Metastatic Renal Cell Carcinoma: Clinical Outcome According to International Metastatic Renal Cell Carcinoma Database Consortium Risk Group. Clin Genitourin Cancer. 2018 Aug;16(4):298-304. doi: 10.1016/j.clgc.2018.04.005. Epub 2018 May 4. PMID 29853320
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Cella D, Michaelson MD, Bushmakin AG, Cappelleri JC, Charbonneau C, Kim ST, Li JZ, Motzer RJ. Health-related quality of life in patients with metastatic renal cell carcinoma treated with sunitinib vs interferon-alpha in a phase III trial: final results and geographical analysis. Br J Cancer. 2010 Feb 16;102(4):658-64. doi: 10.1038/sj.bjc.6605552. Epub 2010 Jan 26. PMID 20104222
- [Derived] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181034&StudyName=SU011248%20Versus%20Interferon-Alfa%20As%20First-Line%20Systemic%20Therapy%20For%20Patients%20With%20Metastatic%20Renal%20Cell%20Carcinoma%20%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 101 medical centers took part in the study between 10 August 2004 and 19 September 2008.
Pre-assignment Details: Subjects were to be followed until survival data was mature (median duration of follow-up: 123 weeks).
Groups:
- SU011248: 50 mg taken orally once a day for 4 weeks followed by a 2-week off treatment cycle to form a 6-week treatment cycle. Intra-subject dose reduction to 37.5 mg/day and 25 mg/day was allowed depending on type and severity of toxicity encountered.
- IFN-α: Subcutaneous (SC) injection in 6-week cycles on 3 non-consecutive days per week; 3 million units (MU) per dose Week 1; 6 MU per dose Week 2; 9 MU per dose Week 3 until completion of therapy or development of toxicity.
Period: Overall Study
Arm/Group | SU011248 | IFN-α
Started | 375 | 375
Received Treatment | 375 | 360 (15 subjects randomized to IFN-α discontinued before receiving their first dose of study medication.)
Completed | 0 | 0 (Discontinuation crossover subjects: AEs 5,consent withdrawn 2, lack efficacy 13, sponsor decision 5.)
Not Completed | 375 | 375
Not completed — Adverse Event | 76 | 86
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 22 | 24
Not completed — Lack of Efficacy | 240 | 219
Not completed — Decision of sponsor | 32 | 4
Not completed — Randomized: did not take study drug | 0 | 15
Not completed — Completed on marketed sunitinub | 3 | 0
Not completed — Crossover to SU011248 | 0 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SU011248 | IFN-α | Total
Number analyzed (Participants) | 375 | 375 | 750
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 223 | 252 | 475
  >=65 years | 152 | 123 | 275
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 106 | 214
  Male | 267 | 269 | 536

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), Core Radiology Assessment
Description: Progression-free survival (PFS) = time from randomization to first documentation of objective tumor progression or to death due to any cause, whichever occured first. If tumor progression data included more than 1 date, the first date was used. PFS = first event date minus the date of randomization + 1. On study included treatment plus 28-day follow-up periods.
Time Frame: Day 28 of each 6-week cycle: duration of treatment phase
Population: Intent to treat (ITT) population: all patients who were randomized, with study drug assignment designated according to initial randomization, regardless of whether patients received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
weeks | 48.3 [46.4 to 58.3] | 22.1 [17.1 to 24.0]
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Unstratified analysis: Hazard Ratio (SU011248 vs IFN-α). Progression-free survival (PFS) was assessed in each treatment arm using the Kaplan-Meier method; Test type: Superiority or Other; p < 0.0001, Log Rank — p-value from 2-sided, unstratified test; Hazard Ratio (HR) = 0.5268, 95% CI 2-sided [0.4316 to 0.6430] — Assuming proportional hazards, a hazard ratio les than 1 indicates a reduction in hazard rate in favor of SU011248; a hazard ratio greater than 1 indicates a reduction in favor of IFN-a
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Stratified analysis: Hazard Ratio (SU011248 vs IFN-a); Test type: Superiority or Other; p < .00001, Log Rank — p-value is from 2-sided, stratified test. Stratification factors were: Lactic Dehydrogenase (LDH) > or <= 1.5 x upper limit of normal, Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, and absence or presence of prior nephrectomy; Hazard Ratio (HR) = 0.5136, 95% CI 2-sided [0.4196 to 0.6288] — Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of SU011248: a hazard ratio greater than 1 indicates a reduction in favor of IFN-a

2. Secondary Outcome: Objective Response, Core Radiology Assessment
Description: Objective response (OR) = the number of patients with confirmed complete response (CR) and confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, relative to all randomized patients. CR was defined as the disappearance of all target lesions. PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Confirmed responses (CR or PR) = those that persisted on repeat imaging study >= 4 weeks after initial documentation of response.
Time Frame: Day 28 of each 6-week cycle: duration of treatment phase
Population: ITT
Measure: Number; unit: participants
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
participants | 145 | 29
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Test type: Superiority or Other; p < 0.001, Chi-squared; treatment difference = 30.93, 95% CI 2-sided [25.31 to 36.56] — 95% confidence interval was calculated based on a normal distribution

3. Secondary Outcome: Objective Response, Investigator's Assessment
Description: Objective response (OR) = the number of patients with confirmed complete response (CR) and confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, relative to all randomized patients. CR was defined as the disappearance of all target lesions. PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Confirmed responses = those that persist on repeat imaging study >= 4 weeks after initial documentation of response.
Time Frame: Day 28 of each 6-week cycle: duration of treatment phase
Population: ITT
Measure: Number; unit: participants
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
participants | 171 | 45
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Test type: Superiority or Other; p < 0.001, Chi-squared; treatment difference = 33.66, 95% CI 2-sided [27.62 to 39.69] — 95% confidence interval was calculated based on a normal distribution

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) = time from date of randomization to date of death due to any cause. For patients not expiring, survival time was censored at the last date they were known to be alive. Patients lacking data beyond randomization had their survival times censored at the date of randomization with a duration of 1 day.
Time Frame: Clinic visit or telephone contact every 2 months until death
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
weeks | 114.6 [100.1 to 142.9] | 94.9 [77.7 to 117.0]
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Unstratified analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p = 0.0510, Log Rank — p-value is from 2-sided, unstratified tests; Hazard Ratio (HR) = 0.8209, 95% CI 2-sided [0.6730 to 1.0013] — Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of SU011248; a hazard ratio greater than 1 indicates a reduction in hazard rate in favor of IFN-a
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Unstratified analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p = 0.0128, Wilcoxon (Mann-Whitney) — p-value is from 2-sided, unstratified tests; Hazard Ratio (HR) = 0.8209, 95% CI 2-sided [0.6730 to 1.0013] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Stratified analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p = 0.0490, Log Rank — p-value is from 2-sided, stratified tests. Stratification factors were: Lactic Dehydrogenase (LDH) > or <= 1.5 x upper limit of normal, Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, and absence or presence of prior nephrectomy; Hazard Ratio (HR) = 0.8179, 95% CI 2-sided [0.6692 to 0.9995] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to Tumor Progression (TTP), Core Radiology Assessment
Description: TTP = time from randomization to first documentation of objective tumor progression. TTP data were censored on the day following the date of last on treatment (including 28 day follow-up period) tumor assessment documenting absence of progressive disease for subjects who did not have objective tumor progression while on treatment or who were given anti-tumor treatment other than study treatment prior to documentation of objective tumor progression. Subjects with no tumor assessments after randomization had TTP censored on the date of randomization with a duration of 1 day.
Time Frame: Randomization to first documentation of tumor progression: duration of treatment phase
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
weeks | 49.1 [46.6 to 59.1] | 22.4 [21.9 to 31.3]
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Unstratified Analysis: Hazard Ratio (SU011248 vs IFN-a); Test type: Superiority or Other; p < 0.0001, Log Rank — p-value is from 2-sided, unstratified test; Hazard Ratio (HR) = 0.5332, 95% CI 2-sided [0.4345 to 0.6544] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Stratified Analysis: Hazard Ratio (SU011248 vs IFN-a); Test type: Superiority or Other; p < .00001, Log Rank — p-value is from 2-sided, stratified test. Stratification factors are: Lactic Dehydrogenase (LDH) > or <= 1.5 x upper limit of normal, Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, and absence or presence of prior nephrectomy; Hazard Ratio (HR) = 0.5160, 95% CI 2-sided [0.4191 to 0.6352] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Time to Tumor Progression (TTP), Investigator's Assessment
Description: TTP = time from randomization to first documentation of objective tumor progression. TTP data were censored on the day following the date of last on treatment (including 28 day follow-up period) tumor assessment documenting absence of progressive disease for subjects who did not have objective tumor progression while on treatment or who were given anti-tumor treatment other than the study treatment prior to documentation of objective tumor progression. Subjects with no tumor assessments after randomization had TTP censored on the date of randomization with a duration of 1 day.
Time Frame: Randomization to first documentation of tumor progression: duration of treatment phase
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
weeks | 49.0 [46.4 to 59.1] | 22.3 [17.3 to 31.6]
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Unstratified Analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p < 0.0001, Log Rank — p-value is from 2-sided, unstratified test; Hazard Ratio (HR) = 0.5454, 95% CI 2-sided [0.4558 to 0.6526] — Assuming proportional hazards, a hazard ratio < 1 indicates a reduction in hazard rate in favor of SU011248; a hazard ratio > 1 indicates a reduction in hazard rate in favor of IFN-a
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Stratified Analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p < .00001, Log Rank — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.5417, 95% CI 2-sided [0.4519 to 0.6492] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Duration of Response (DR), Core Radiology Assessement
Description: Duration of response (DR) = time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause. DR data were censored on the day following the date of the last on treatment (including 28 day follow-up period) tumor assessment documenting absence of progressive disease for subjects without objective tumor progression who did not die due to any cause while on treatment or who were given anti-tumor treatment other than study treatment prior to observing tumor progression.
Time Frame: Day 28 of each cycle: duraton of treatment phase
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 71 | 9
weeks | 52.9 [46.1 to 60.1] | 64.9 [41.9 to 82.0]

8. Secondary Outcome: Duration of Response (DR), Investigator's Assessment
Description: Duration of response (DR) = time from the first documentation of objective tumor response to the first documentaion of objective tumor progression or to death due to any cause. DR data were censored on the day following the date of the last on treatment (including 28 day follow-up period) tumor assessment documenting absence of progressive disease for subjects without objective tumor progression who did not die due to any cause while on treatment or who were given anti-tumor treatment other than study treatment prior to observing tumor progression.
Time Frame: Day 28 of each cycle: duration of treatment phase
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 122 | 23
weeks | 56.3 [48.4 to 64.9] | 48.1 [42.1 to 120.1]

9. Secondary Outcome: FACT-Kidney Symptom Index-Disease Related Symptoms (FKSI-DRS) Subscale
Description: FACT-Kidney Symptom Index-Disease Related Symptoms (FKSI-DRS) subscale of the FKSI to measure advanced kidney cancer disease related symptoms. Includes 9 items: lack of energy, pain, losing weight, bone pain, fatigue, short of breath, coughing, bothered by fevers, and hematuria. Each question was answered on a five-point Likert-type scale ranging from 0 (not at all) to 4 (very much). Score = the sum score of the item scores in the subscale; total range: 0 to 36. A score greater than 0 indicates the difference favored sunitinib.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; summary of FKSI-DRS questionnaire results by treatment; N=number of subjects with evaluable data; n = number of subjects with evaluable data at observation, SU011248 and INF-α treatment groups, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=368, 351) | 29.74 (5.244) | 29.55 (5.026)
  Cycle 1 Day 28 (n=348, 317) | 27.73 (5.080) [29.000 to 29.663] | 26.68 (5.195) [27.011 to 27.782]
  Cycle 2 Day 1 (n=327, 246) | 29.66 (4.778) [29.019 to 29.667] | 27.59 (4.908) [27.016 to 27.775]
  Cycle 2 Day 28 (n= 315, 237) | 28.49 (4.748) [29.051 to 29.677] | 27.22 (4.988) [27.019 to 27.769]
  Cycle 3 Day 1 (n=294, 198) | 29.93 (4.679) [29.068 to 29.684] | 28.20 (4.452) [27.017 to 27.770]
  Cycle 3 Day 28 (n=285, 195) | 28.72 (4.756) [29.095 to 29.698] | 27.81 (5.040) [27.006 to 27.778]
  Cycle 4 Day 1 (n=272, 151) | 30.25 (4.498) | 28.85 (4.821)
  Cycle 4 Day 28 (n=264, 142) | 29.43 (4.389) | 28.30 (5.071)
  Cycle 5 Day 1 (n=248, 119 ) | 30.87 (3.948) | 28.57 (4.925)
  Cycle 5 Day 28 (n=242, 109) | 29.43 (4.280) | 28.37 (4.726)
  Cycle 6 Day 1 (n=240, 99) | 30.80 (4.214) | 29.12 (4.428)
  Cycle 6 Day 28 (n=223, 99) | 29.62 (4.288) | 28.44 (4.957)
  Cycle 7 Day 1 (n=208, 79) | 30.93 (4.002) | 28.99 (4.974)
  Cycle 7 Day 28 (n=203, 75 ) | 29.73 (4.417) | 28.50 (4.556)
  Cycle 8 Day 1 (n=192, 68) | 31.03 (3.649) | 28.76 (4.847)
  Cycle 8 Day 28 (n=190, 62) | 29.76 (4.096) | 28.67 (4.491)
  Cycle 9 Day 1 (n=172, 51) | 31.24 (3.560) | 29.86 (4.247)
  Cycle 9 Day 28 (n=166, 46) | 29.72 (4.245) | 29.36 (4.418)
  Cycle 10 Day 1 (n=161, 50) | 30.73 (3.820) | 29.43 (4.455)
  Cycle 10 Day 28 (n=155, 46) | 29.78 (4.034) | 29.03 (4.980)
  Cycle 11 Day 1 (n=138, 35) | 30.72 (4.018) | 29.89 (4.006)
  Cycle 11 Day 28 (n=141, 33) | 29.34 (4.117) | 29.24 (5.014)
  Cycle 12 Day 1 (n=132, 31) | 30.76 (4.108) | 29.54 (5.607)
  Cycle 12 Day 28 (n=128, 31) | 29.63 (4.362) | 29.48 (4.774)
  Cycle 13 Day 1 (113, 27) | 30.58 (4.354) | 29.81 (4.923)
  Cycle 13 Day 28 (n=114, 27) | 29.30 (4.424) | 29.63 (4.550)
  Cycle 14 Day 1 (n=114, 26) | 30.58 (4.179) | 29.35 (4.664)
  Cycle 14 Day 28 (n=105, 25) | 28.94 (4.771) | 29.23 (5.502)
  Cycle 15 Day 1 (n=100, 22) | 30.87 (4.075) | 29.18 (5.917)
  Cycle 15 Day 28 (n=94, 20) | 29.26 (4.320) | 28.89 (5.676)
  Cycle 16 Day 1 (n=96, 19) | 30.63 (3.786) | 27.79 (5.760)
  Cycle 16 Day 28 (n=90, 18) | 29.51 (4.302) | 28.28 (6.267)
  Cycle 17 Day 1 (n=85, 17) | 30.69 (4.132) | 29.26 (5.434)
  Cycle 17 Day 28 (n=81, 14) | 29.73 (4.155) | 27.94 (7.519)
  Cycle 18 Day 1 (n=80, 12) | 30.24 (4.091) | 28.83 (7.209)
  Cycle 18 Day 28 (n=70, 11) | 29.15 (4.358) | 28.73 (6.973)
  Cycle 19 Day 1 (n=71, 11) | 30.11 (4.528) | 29.64 (7.061)
  Cycle 19 Day 28 (n=61, 10) | 29.48 (4.678) | 28.65 (8.131)
  Cycle 20 Day 1 (n=65, 9) | 31.07 (4.073) | 28.44 (8.048)
  Cycle 20 Day 28 (n=53, 9) | 29.44 (4.210) | 29.22 (7.694)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index-Disease Related Symptoms (FKSI-DRS) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.913, 95% CI 2-sided [1.376 to 2.450]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Difference in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.935, 95% CI 2-sided [1.421 to 2.449]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Difference in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.948, 95% CI 2-sided [1.443 to 2.452]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.970, 95% CI 2-sided [1.476 to 2.464]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.983, 95% CI 2-sided [1.491 to 2.475]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.005, 95% CI 2-sided [1.510 to 2.501]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.018, 95% CI 2-sided [1.517 to 2.519]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.040, 95% CI 2-sided [1.522 to 2.559]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.053, 95% CI 2-sided [1.522 to 2.584]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.075, 95% CI 2-sided [1.515 to 2.635]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.088, 95% CI 2-sided [1.509 to 2.667]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.110, 95% CI 2-sided [1.494 to 2.727]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.123, 95% CI 2-sided [1.483 to 2.763]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.146, 95% CI 2-sided [1.461 to 2.830]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Median Difference (Final Values) = 2.158, 95% CI 2-sided [1.447 to 2.869]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.181, 95% CI 2-sided [1.420 to 2.941]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.193, 95% CI 2-sided [1.404 to 2.983]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.216, 95% CI 2-sided [1.373 to 3.059]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.228, 95% CI 2-sided [1.355 to 3.102]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.251, 95% CI 2-sided [1.321 to 3.180]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.263, 95% CI 2-sided [1.302 to 3.225]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.286, 95% CI 2-sided [1.266 to 3.305]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.298, 95% CI 2-sided [1.246 to 3.351]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.321, 95% CI 2-sided [1.209 to 3.433]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.333, 95% CI 2-sided [1.188 to 3.479]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.356, 95% CI 2-sided [1.150 to 3.562]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 2.369, 95% CI 2-sided [1.128 to 3.609]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 2.391, 95% CI 2-sided [1.089 to 3.693]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 2.404, 95% CI 2-sided [1.067 to 3.740]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 2.426, 95% CI 2-sided [1.027 to 3.825]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = 2.439, 95% CI [1.005 to 3.872]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mean Difference (Final Values) = 2.461, 95% CI 2-sided [0.964 to 3.958]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = 2.474, 95% CI 2-sided [0.942 to 4.006]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = 2.496, 95% CI 2-sided [0.901 to 4.092]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; Mean Difference (Final Values) = 2.509, 95% CI 2-sided [0.878 to 4.140]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; Mean Difference (Final Values) = 2.531, 95% CI 2-sided [0.836 to 4.226]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis; Mean Difference (Final Values) = 2.544, 95% CI 2-sided [0.813 to 4.274]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; Mean Difference (Final Values) = 2.566, 95% CI 2-sided [0.772 to 4.361]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis; Mean Difference (Final Values) = 2.579, 95% CI 2-sided [0.748 to 4.410]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FKSI-DRS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; Mean Difference (Final Values) = 2.602, 95% CI 2-sided [0.706 to 4.497]

10. Secondary Outcome: FACT-Kidney Symptom Index (FKSI) Subscale
Description: FACT-Kidney Symptom Index (FKSI) subscale designed to be a stand-alone instrument to measure symptoms and quality of life in patients with advanced kidney cancer. Contains 15 questions; some questions overlap with the FACT-G questions. Each question was answered on a five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Total FKSI score = sum score of the 15 item scores; total range: 0 - 60; 0 (most severe symptoms and concerns) to 60 (no symptoms or concerns).
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=369, 351) | 46.45 (8.464) | 46.09 (8.701)
  Cycle 1 Day 28 (n=348, 317) | 42.71 (8.959) | 40.93 (9.292)
  Cycle 2 Day 1 (n=327, 246) | 45.98 (8.401) | 42.33 (8.733)
  Cycle 2 Day 28 (n=315, 238) | 43.75 (8.607) | 42.01 (8.659)
  Cycle 3 Day 1 (n=294, 198) | 46.60 (8.263) | 43.64 (7.983)
  Cycle 3 Day 28 (n=285, 195) | 44.01 (8.529) | 43.13 (8.925)
  Cycle 4 Day 1 (n=272, 151) | 46.99 (8.041) | 44.78 (8.328)
  Cycle 4 Day 28 (n=264, 142) | 45.08 (8.017) | 44.03 (8.913)
  Cycle 5 Day 1 (n=248, 119) | 47.99 (7.313) | 44.82 (8.293)
  Cycle 5 Day 28 (n=242, 109) | 44.99 (7.768) | 44.41 (8.318)
  Cycle 6 Day 1 (n=240, 99) | 47.61 (7.860) | 45.38 (7.995)
  Cycle 6 Day 28 (n=223, 99) | 45.40 (7.840) | 44.07 (9.003)
  Cycle 7 Day 1 (n=208, 79) | 47.84 (7.303) | 45.09 (9.061)
  Cycle 7 Day 28 (n=203, 75) | 45.39 (8.013) | 44.65 (8.082)
  Cycle 8 Day 1 (n=192, 68) | 48.24 (6.818) | 45.38 (8.597)
  Cycle 8 Day 28 (n=190, 62) | 45.83 (7.589) | 45.10 (8.197)
  Cycle 9 Day 1 (n=172, 51) | 48.31 (6.971) | 46.88 (7.901)
  Cycle 9 Day 28 (n=166, 46) | 45.79 (7.969) | 46.16 (8.133)
  Cycle 10 Day 1 (n=161, 50) | 47.90 (6.993) | 46.22 (7.778)
  Cycle 10 Day 28 (n=155, 46) | 45.70 (7.372) | 45.16 (8.961)
  Cycle 11 Day 1 (n=138, 35) | 47.90 (6.988) | 46.26 (7.398)
  Cycle 11 Day 28 (n=141, 33) | 45.28 (7.330) | 45.46 (8.920)
  Cycle 12 Day 1 (n=132, 31) | 47.90 (7.458) | 46.08 (9.456)
  Cycle 12 Day 28 (n=128, 31) | 45.67 (7.696) | 46.00 (8.802)
  Cycle 13 Day 1 (n=113, 27) | 48.02 (7.723) | 46.25 (8.833)
  Cycle 13 Day 28 (n=114, 27) | 45.65 (7.659) | 45.84 (9.095)
  Cycle 14 Day 1 (n=114, 26) | 47.90 (7.370) | 46.08 (8.621)
  Cycle 14 Day 28 (n=105, 25) | 45.10 (8.641) | 46.10 (9.650)
  Cycle 15 Day 1 (n=100, 22) | 48.26 (7.663) | 45.62 (9.715)
  Cycle 15 Day 28 (n=94, 20) | 45.37 (8.040) | 45.30 (9.776)
  Cycle 16 Day 1 (n=96, 19) | 47.75 (7.063) | 43.64 (10.688)
  Cycle 16 Day 28 (n=90, 18) | 45.95 (7.625) | 43.46 (10.549)
  Cycle 17 Day 1 (n=85, 17) | 48.07 (7.641) | 45.59 (10.302)
  Cycle 17 Day 28 (n=81, 14) | 46.27 (8.016) | 43.64 (11.693)
  Cycle 18 Day 1 (n=80, 12) | 47.47 (7.598) | 44.92 (12.391)
  Cycle 18 Day 28 (n=70, 11) | 45.36 (7.585) | 45.27 (11.909)
  Cycle 19 Day 1 (n=71, 11) | 47.70 (7.671) | 46.64 (12.808)
  Cycle 19 Day 28 (n=61, 10) | 46.07 (8.442) | 44.47 (14.476)
  Cycle 20 Day 1 (n=65, 9) | 48.88 (7.133) | 45.00 (13.811)
  Cycle 20 Day 28 (n=53, 9) | 46.26 (8.065) | 46.00 (13.266)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.165, 95% CI 2-sided [2.234 to 4.095]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.205, 95% CI 2-sided [2.318 to 4.092]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.228, 95% CI 2-sided [2.358 to 4.097]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.268, 95% CI 2-sided [2.418 to 4.119]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.291, 95% CI 2-sided [2.443 to 4.139]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.331, 95% CI 2-sided [2.474 to 4.189]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.354, 95% CI [2.484 to 4.224]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.395, 95% CI 2-sided [2.489 to 4.300]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.417, 95% CI 2-sided [2.486 to 4.348]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.458, 95% CI 2-sided [2.469 to 4.446]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.480, 95% CI 2-sided [2.455 to 4.505]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.521, 95% CI 2-sided [2.422 to 4.620]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.543, 95% CI 2-sided [2.399 to 4.687]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.584, 95% CI [2.354 to 4.814]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.606, 95% CI 2-sided [2.326 to 4.887]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.647, 95% CI 2-sided [2.272 to 5.022]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.669, 95% CI 2-sided [2.240 to 5.099]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.710, 95% CI 2-sided [2.180 to 5.240]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.733, 95% CI 2-sided [2.145 to 5.320]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.773, 95% CI 2-sided [2.080 to 5.466]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.796, 95% CI 2-sided [2.043 to 5.548]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.836, 95% CI 2-sided [1.975 to 5.698]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.859, 95% CI 2-sided [1.936 to 5.781]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 3.899, 95% CI 2-sided [1.866 to 5.933]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 3.922, 95% CI 2-sided [1.826 to 6.018]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 3.962, 95% CI 2-sided [1.753 to 6.172]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 3.985, 95% CI [1.712 to 6.258]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 4.026, 95% CI 2-sided [1.638 to 6.413]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Mean Difference (Final Values) = 4.048, 95% CI 2-sided [1.597 to 6.500]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 4.089, 95% CI 2-sided [1.521 to 6.656]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = 4.111, 95% CI 2-sided [1.479 to 6.743]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; Mean Difference (Final Values) = 4.152, 95% CI 2-sided [1.403 to 6.901]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; Mean Difference (Final Values) = 4.174, 95% CI [1.360 to 6.988]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis; Mean Difference (Final Values) = 4.215, 95% CI 2-sided [1.283 to 7.147]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; Mean Difference (Final Values) = 4.237, 95% CI 2-sided [1.240 to 7.235]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; Mean Difference (Final Values) = 4.278, 95% CI 2-sided [1.162 to 7.394]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis; Mean Difference (Final Values) = 4.300, 95% CI 2-sided [1.119 to 7.482]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis; Mean Difference (Final Values) = 4.341, 95% CI 2-sided [1.041 to 7.642]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0111, Mixed Models Analysis; Mean Difference (Final Values) = 4.364, 95% CI 2-sided [0.997 to 7.730]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-Kidney Symptom Index (FKSI) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis; Mean Difference (Final Values) = 4.404, 95% CI 2-sided [0.918 to 7.890]

11. Primary Outcome: Progression-Free Survival (PFS), Investigator's Assessment
Description: Progression-free survival = time from randomization to first documentation of objective tumor progression or to death due to any cause, whichever occured first. PFS = first event date minus the date of randomization + 1). On study included treatment plus 28-day follow-up periods.
Time Frame: Day 28 of each 6-week cycle: duration of treatment phase
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
weeks | 47.7 [46.3 to 58.1] | 22.1 [16.7 to 27.4]
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Unstratified analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p < 0.0001, Log Rank — p-value is from 2-sided, unstratified test; Hazard Ratio (HR) = 0.5404, 95% CI 2-sided [0.4532 to 0.6444] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Stratified analysis: Hazard Ratio (SU011248 vs IFN-α); Test type: Superiority or Other; p < .00001, Log Rank — [p-value comment as in outcome 5, analysis 2]; Hazard Ratio (HR) = 0.5418, 95% CI 2-sided [0.4536 to 0.6473] — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Functional Assessment of Cancer Therapy-General (FACT-G): core questionnaire of the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system that has been validated in a variety of cancer populations. 27 questions grouped into 4 domains that measure a patient's physical, functional, social and family, and emotional well-being. Five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Score = sum score of item scores in the subscale; total range: 0 to 108 with higher score indicating better quality of life.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=368, 346) | 82.30 (15.213) | 81.22 (16.030)
  Cycle 1 Day 28 (n=345, 316) | 78.75 (15.702) | 74.91 (18.374)
  Cycle 2 Day 1 (n=328, 247) | 82.88 (15.733) | 77.02 (16.670)
  Cycle 2 Day 28 (n=314, 237) | 80.51 (16.229) | 77.05 (17.468)
  Cycle 3 Day 1 (n=293, 199) | 84.24 (16.121) | 79.35 (16.862)
  Cycle 3 Day 28 (n=285, 193) | 80.59 (16.144) | 78.42 (17.836)
  Cycle 4 Day 1 (n=269, 149) | 85.32 (14.723) | 80.86 (16.477)
  Cycle 4 Day 28 (n=263, 142) | 82.08 (15.147) | 80.46 (17.136)
  Cycle 5 Day 1 (n=247, 119) | 86.40 (14.019) | 81.96 (15.286)
  Cycle 5 Day 28 (n=240, 106) | 82.23 (15.124) | 80.60 (15.527)
  Cycle 6 Day 1 (n=238, 98) | 84.90 (15.189) | 81.97 (15.918)
  Cycle 6 Day 28 (n=222, 97) | 82.54 (15.338) | 79.70 (16.686)
  Cycle 7 Day 1 (n=206, 78) | 85.01 (15.118) | 80.39 (17.811)
  Cycle 7 Day 28 (n=200, 75) | 82.16 (16.207) | 81.06 (16.701)
  Cycle 8 Day 1 (n=192, 66) | 86.83 (13.456) | 81.25 (17.179)
  Cycle 8 Day 28 (n=189, 61) | 83.05 (14.699) | 81.31 (16.700)
  Cycle 9 Day 1 (n=170, 51) | 85.81 (14.865) | 84.50 (16.174)
  Cycle 9 Day 28 (n=166, 46) | 82.71 (15.276) | 83.14 (17.067)
  Cycle 10 Day 1 (n=158, 49) | 85.32 (14.500) | 84.03 (16.559)
  Cycle 10 Day 28 (n=150, 45) | 82.14 (15.193) | 81.79 (17.994)
  Cycle 11 Day 1 (n=134, 35) | 84.75 (14.791) | 81.60 (16.729)
  Cycle 11 Day 28 (n=139, 32) | 81.91 (14.865) | 80.20 (19.213)
  Cycle 12 Day 1 (n=130, 29) | 85.31 (15.181) | 80.99 (20.219)
  Cycle 12 Day 28 (n=126, 31) | 82.43 (15.152) | 81.73 (18.745)
  Cycle 13 Day 1 (n=113, 27) | 85.50 (15.209) | 81.18 (20.198)
  Cycle 13 Day 28 (n=114, 27) | 83.61 (14.445) | 80.67 (18.678)
  Cycle 14 Day 1 (n=112, 26) | 85.24 (14.398) | 81.22 (17.506)
  Cycle 14 Day 28 (n=107, 24) | 82.34 (16.300) | 81.57 (20.188)
  Cycle 15 Day 1 (n=101, 20) | 86.24 (14.742) | 81.66 (18.326)
  Cycle 15 Day 28 (n=96, 20) | 82.64 (15.722) | 80.88 (18.913)
  Cycle 16 Day 1 (n=94, 19) | 84.77 (14.741) | 78.20 (18.994)
  Cycle 16 Day 28 (n=89, 18) | 83.38 (15.481) | 78.38 (19.749)
  Cycle 17 Day 1 (n=84, 16) | 86.78 (14.800) | 81.80 (20.161)
  Cycle 17 Day 28 (n=80, 14) | 84.42 (15.106) | 78.96 (21.571)
  Cycle 18 Day 1 (n=79, 12) | 85.74 (14.987) | 82.24 (23.763)
  Cycle 18 Day 28 (n=70, 11) | 83.51 (14.831) | 82.27 (21.950)
  Cycle 19 Day 1 (n=71, 11) | 87.16 (14.245) | 82.48 (24.198)
  Cycle 19 Day 28 (n=61, 10) | 84.54 (16.679) | 79.63 (27.938)
  Cycle 20 Day 1 (n=63, 9) | 87.96 (14.441) | 81.70 (27.018)
  Cycle 20 Day 28 (n=52, 8) | 84.62 (16.257) | 79.54 (26.109)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Functional Assessment of Cancer Therapy-General (FACT-G) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.486, 95% CI 2-sided [3.852 to 7.119]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.535, 95% CI 2-sided [3.955 to 7.115]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.562, 95% CI 2-sided [4.000 to 7.124]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.611, 95% CI 2-sided [4.061 to 7.162]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.639, 95% CI 2-sided [4.083 to 7.195]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.688, 95% CI 2-sided [4.100 to 7.276]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.715, 95% CI 2-sided [4.098 to 7.333]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.764, 95% CI 2-sided [4.075 to 7.454]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.792, 95% CI 2-sided [4.053 to 7.531]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.841, 95% CI 2-sided [3.998 to 7.684]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.868, 95% CI 2-sided [3.960 to 7.777]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.917, 95% CI 2-sided [3.880 to 7.955]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.945, 95% CI 2-sided [3.830 to 8.060]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.994, 95% CI 2-sided [3.731 to 8.257]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.021, 95% CI 2-sided [3.672 to 8.370]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.071, 95% CI 2-sided [3.560 to 8.581]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.098, 95% CI 2-sided [3.495 to 8.701]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.147, 95% CI 2-sided [3.373 to 8.921]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.174, 95% CI 2-sided [3.303 to 9.045]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.224, 95% CI 2-sided [3.174 to 9.273]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 6.251, 95% CI 2-sided [3.101 to 9.401]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 6.300, 95% CI 2-sided [2.966 to 9.634]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 6.327, 95% CI 2-sided [2.890 to 9.765]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 6.377, 95% CI 2-sided [2.751 to 10.002]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 6.404, 95% CI 2-sided [2.673 to 10.135]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mean Difference (Final Values) = 6.453, 95% CI 2-sided [2.530 to 10.376]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = 6.480, 95% CI 2-sided [2.451 to 10.510]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; Mean Difference (Final Values) = 6.530, 95% CI 2-sided [2.306 to 10.754]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis; Mean Difference (Final Values) = 6.557, 95% CI 2-sided [2.224 to 10.889]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0043, Mixed Models Analysis; Mean Difference (Final Values) = 6.606, 95% CI 2-sided [2.077 to 11.135]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; Mean Difference (Final Values) = 6.634, 95% CI 2-sided [1.995 to 11.272]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0068, Mixed Models Analysis; Mean Difference (Final Values) = 6.683, 95% CI 2-sided [1.847 to 11.519]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0079, Mixed Models Analysis; Mean Difference (Final Values) = 6.710, 95% CI 2-sided [1.764 to 11.657]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0100, Mixed Models Analysis; Mean Difference (Final Values) = 6.759, 95% CI 2-sided [1.613 to 11.905]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0114, Mixed Models Analysis; Mean Difference (Final Values) = 6.787, 95% CI 2-sided [1.530 to 12.043]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0141, Mixed Models Analysis; Mean Difference (Final Values) = 6.836, 95% CI 2-sided [1.378 to 12.293]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0157, Mixed Models Analysis; Mean Difference (Final Values) = 6.863, 95% CI 2-sided [1.294 to 12.432]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0189, Mixed Models Analysis; Mean Difference (Final Values) = 6.912, 95% CI 2-sided [1.142 to 12.683]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0208, Mixed Models Analysis; Mean Difference (Final Values) = 6.940, 95% CI 2-sided [1.057 to 12.822]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0244, Mixed Models Analysis; Mean Difference (Final Values) = 6.989, 95% CI 2-sided [0.904 to 13.074]

13. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G): Physical Well Being (PWB) Subscale
Description: Physical well-being (PWB) subscale of the Functional Assessment of Cancer Therapy-General (FACT-G). Each question was answered on a five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Score = the sum score of the item scores in the subscale; range: 0 to 28; lower score indicates better physical well-being.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=369, 348) | 23.14 (5.209) | 22.70 (5.224)
  Cycle 1 Day 28 (n=348, 318) | 19.43 (6.052) | 18.85 (6.168)
  Cycle 2 Day 1 (n=329, 247) | 22.22 (5.161) | 20.05 (5.499)
  Cycle 2 Day 28 (n=316, 239) | 20.34 (5.654) | 19.84 (5.706)
  Cycle 3 Day 1 (n=294, 200) | 22.45 (5.123) | 20.87 (5.281)
  Cycle 3 Day 28 (n=286, 195) | 20.18 (5.650) | 20.63 (5.395)
  Cycle 4 Day 1 (n=270, 150) | 22.72 (4.641) | 21.56 (4.581)
  Cycle 4 Day 28 (n=264, 142) | 21.00 (5.120) | 21.31 (5.110)
  Cycle 5 Day 1 (n=248, 120) | 23.24 (4.143) | 21.84 (4.567)
  Cycle 5 Day 28 (n=241, 106) | 20.91 (5.062) | 21.23 (4.867)
  Cycle 6 Day 1 (n=239, 99) | 22.99 (4.385) | 21.70 (4.761)
  Cycle 6 Day 28 (n=224, 97) | 21.22 (5.070) | 20.96 (5.384)
  Cycle 7 Day 1 (n=207, 79) | 23.05 (4.414) | 21.67 (4.964)
  Cycle 7 Day 28 (n=201, 75) | 21.22 (5.250) | 21.66 (4.595)
  Cycle 8 Day 1 (n=193, 67) | 23.58 (3.715) | 21.94 (4.870)
  Cycle 8 Day 28 (n=189, 61) | 21.51 (4.666) | 21.40 (4.910)
  Cycle 9 Day 1 (n=172, 51) | 23.41 (4.071) | 22.58 (4.367)
  Cycle 9 Day 28 (n=166, 46) | 21.29 (5.068) | 22.38 (4.400)
  Cycle 10 Day 1 (n=159, 49) | 22.94 (4.053) | 22.60 (4.124)
  Cycle 10 Day 28 (n=151, 46) | 21.21 (4.848) | 21.83 (5.165)
  Cycle 11 Day 1 (n=135, 35) | 23.16 (4.069) | 22.23 (4.194)
  Cycle 11 Day 28 (n=140, 32) | 20.98 (4.597) | 21.88 (5.173)
  Cycle 12 Day 1 (n=131, 30) | 23.03 (4.291) | 22.60 (5.236)
  Cycle 12 Day 28 (n=127, 31) | 20.87 (4.721) | 21.90 (4.867)
  Cycle 13 Day 1 (n=114, 27) | 23.05 (4.281) | 21.99 (5.187)
  Cycle 13 Day 28 (n=114, 27) | 21.26 (4.623) | 21.80 (5.369)
  Cycle 14 Day 1 (n=112, 26) | 23.02 (4.401) | 22.05 (4.906)
  Cycle 14 Day 28 (n=107, 24) | 20.80 (5.310) | 22.75 (4.875)
  Cycle 15 Day 1 (n=101, 21) | 23.26 (4.475) | 22.33 (5.173)
  Cycle 15 Day 28 (n=96, 20) | 20.95 (4.978) | 22.07 (4.908)
  Cycle 16 Day 1 (n=94, 19) | 22.60 (4.337) | 20.63 (6.125)
  Cycle 16 Day 28 (n=90, 18) | 21.31 (4.939) | 21.42 (6.194)
  Cycle 17 Day 1 (n=85, 16) | 22.99 (4.513) | 21.81 (5.776)
  Cycle 17 Day 28 (n=80, 14) | 21.68 (4.653) | 20.50 (6.757)
  Cycle 18 Day 1 (n=79, 12) | 22.85 (4.388) | 21.83 (6.672)
  Cycle 18 Day 28 (n=70, 11) | 20.89 (5.006) | 22.45 (5.610)
  Cycle 19 Day 1 (n=71, 11) | 23.20 (4.426) | 22.45 (6.773)
  Cycle 19 Day 28 (n=61, 10) | 21.82 (4.696) | 21.60 (7.457)
  Cycle 20 Day 1 (n=63, 9) | 23.68 (4.204) | 21.78 (7.311)
  Cycle 20 Day 28 (n=52, 9) | 21.81 (4.835) | 22.33 (6.423)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Functional Assessment of Cancer Therapy-General (FACT-G) Physical Well Being (PWB) subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.459, 95% CI 2-sided [0.805 to 2.114]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.453, 95% CI 2-sided [0.827 to 2.079]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.450, 95% CI 2-sided [0.837 to 2.063]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.444, 95% CI 2-sided [0.847 to 2.041]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.440, 95% CI 2-sided [0.848 to 2.032]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.434, 95% CI 2-sided [0.844 to 2.024]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.431, 95% CI 2-sided [0.838 to 2.023]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.424, 95% CI 2-sided [0.819 to 2.029]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.421, 95% CI 2-sided [0.805 to 2.037]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.415, 95% CI 2-sided [0.774 to 2.056]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.411, 95% CI 2-sided [0.753 to 2.069]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.405, 95% CI 2-sided [0.711 to 2.099]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.402, 95% CI 2-sided [0.685 to 2.119]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 1.396, 95% CI 2-sided [0.634 to 2.157]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 1.392, 95% CI 2-sided [0.604 to 2.180]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Mean Difference (Final Values) = 1.386, 95% CI 2-sided [0.547 to 2.225]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 1.383, 95% CI 2-sided [0.514 to 2.252]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; Mean Difference (Final Values) = 1.376, 95% CI 2-sided [0.451 to 2.301]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis; Mean Difference (Final Values) = 1.373, 95% CI 2-sided [0.416 to 2.330]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0084, Mixed Models Analysis; Mean Difference (Final Values) = 1.367, 95% CI 2-sided [0.350 to 2.383]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0110, Mixed Models Analysis; Mean Difference (Final Values) = 1.363, 95% CI 2-sided [0.313 to 2.414]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0168, Mixed Models Analysis; Mean Difference (Final Values) = 1.357, 95% CI 2-sided [0.245 to 2.470]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0208, Mixed Models Analysis; Mean Difference (Final Values) = 1.354, 95% CI 2-sided [0.206 to 2.501]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0293, Mixed Models Analysis; Mean Difference (Final Values) = 1.348, 95% CI 2-sided [0.136 to 2.559]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0348, Mixed Models Analysis; Mean Difference (Final Values) = 1.344, 95% CI 2-sided [0.096 to 2.592]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0459, Mixed Models Analysis; Mean Difference (Final Values) = 1.338, 95% CI 2-sided [0.024 to 2.652]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0528, Mixed Models Analysis; Mean Difference (Final Values) = 1.335, 95% CI 2-sided [-0.016 to 2.685]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0663, Mixed Models Analysis; Mean Difference (Final Values) = 1.328, 95% CI 2-sided [-0.090 to 2.746]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0744, Mixed Models Analysis; Mean Difference (Final Values) = 1.325, 95% CI 2-sided [-0.131 to 2.780]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0898, Mixed Models Analysis; Mean Difference (Final Values) = 1.319, 95% CI 2-sided [-0.205 to 2.842]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0988, Mixed Models Analysis; Mean Difference (Final Values) = 1.315, 95% CI 2-sided [-0.246 to 2.877]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1156, Mixed Models Analysis; Mean Difference (Final Values) = 1.309, 95% CI 2-sided [-0.321 to 2.940]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1252, Mixed Models Analysis; Mean Difference (Final Values) = 1.306, 95% CI 2-sided [-0.363 to 2.975]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1429, Mixed Models Analysis; Mean Difference (Final Values) = 1.300, 95% CI 2-sided [-0.439 to 3.038]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1529, Mixed Models Analysis; Mean Difference (Final Values) = 1.296, 95% CI 2-sided [-0.481 to 3.074]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1711, Mixed Models Analysis; Mean Difference (Final Values) = 1.290, 95% CI 2-sided [-0.558 to 3.138]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1813, Mixed Models Analysis; Mean Difference (Final Values) = 1.287, 95% CI 2-sided [-0.600 to 3.173]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1998, Mixed Models Analysis; Mean Difference (Final Values) = 1.280, 95% CI 2-sided [-0.677 to 3.238]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2100, Mixed Models Analysis; Mean Difference (Final Values) = 1.277, 95% CI 2-sided [-0.720 to 3.273]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G PWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2283, Mixed Models Analysis; Mean Difference (Final Values) = 1.271, 95% CI 2-sided [-0.797 to 3.338]

14. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G): Social/Family Well Being (SWB) Subscale
Description: Social/family well-being (SWB)subscale of the Functional Assessment of Cancer Therapy-General (FACT-G). Each question was answered on a five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Score = the sum score of the item scores in the subscale; range: 0 to 28; lower score indicates less social/family well-being.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=370, 349) | 23.14 (4.641) | 22.94 (4.735)
  Cycle 1 Day 28 (n=348, 319) | 23.60 (4.088) | 22.20 (5.076)
  Cycle 2 Day 1 (n=328, 247) | 23.50 (4.344) | 22.31 (5.190)
  Cycle 2 Day 28 (n=315, 238) | 23.40 (4.471) | 22.22 (5.203)
  Cycle 3 Day 1 (n=292, 200) | 23.51 (4.375) | 22.42 (5.011)
  Cycle 3 Day 28 (n=284, 194) | 23.44 (4.369) | 22.12 (5.289)
  Cycle 4 Day 1 (n=269, 150) | 23.73 (4.072) | 22.26 (5.275)
  Cycle 4 Day 28 (n=263, 142) | 23.36 (4.451) | 22.38 (5.198)
  Cycle 5 Day 1 (n=247, 120) | 23.53 (4.334) | 22.35 (5.486)
  Cycle 5 Day 28 (n=241, 107) | 23.68 (4.137) | 22.36 (4.956)
  Cycle 6 Day 1 (n=238, 98) | 23.35 (4.428) | 22.56 (4.678)
  Cycle 6 Day 28 (n=224, 97) | 23.40 (4.393) | 22.33 (4.641)
  Cycle 7 Day 1 (n=207, 79) | 23.29 (4.532) | 22.46 (4.722)
  Cycle 7 Day 28 (n=200, 75) | 23.13 (4.585) | 22.10 (5.286)
  Cycle 8 Day 1 (n=193, 67) | 23.67 (4.225) | 21.95 (5.112)
  Cycle 8 Day 28 (n=189, 61) | 23.26 (4.402) | 22.17 (5.236)
  Cycle 9 Day 1 (n=172, 51) | 23.26 (4.376) | 22.74 (4.826)
  Cycle 9 Day 28 (n=166, 46) | 23.26 (4.395) | 21.96 (5.418)
  Cycle 10 Day 1 (n=158, 49) | 23.08 (4.348) | 22.45 (5.279)
  Cycle 10 Day 28 (n=151, 46) | 23.03 (4.417) | 22.06 (5.065)
  Cycle 11 Day 1 (n=135, 35) | 23.05 (4.521) | 21.51 (5.267)
  Cycle 11 Day 28 (n=140, 32) | 22.71 (4.624) | 21.09 (5.957)
  Cycle 12 Day 1 (n=131, 30) | 23.23 (4.563) | 20.79 (6.007)
  Cycle 12 Day 28 (n=127, 31) | 23.07 (4.586) | 21.25 (5.627)
  Cycle 13 Day 1 (n=114, 27) | 23.15 (4.498) | 20.93 (6.142)
  Cycle 13 Day 28 (n=114, 27) | 23.31 (4.255) | 21.30 (5.491)
  Cycle 14 Day 1 (n=112, 26) | 22.82 (4.647) | 21.51 (5.510)
  Cycle 14 Day 28 (n=107, 24) | 23.24 (4.503) | 20.32 (6.628)
  Cycle 15 Day 1 (n=101, 21) | 23.28 (4.178) | 20.35 (5.986)
  Cycle 15 Day 28 (n=96, 20) | 23.04 (4.312) | 20.23 (6.162)
  Cycle 16 Day 1 (n=94, 19) | 23.11 (4.335) | 21.41 (5.196)
  Cycle 16 Day 28 (n=89, 18) | 23.41 (4.322) | 21.52 (5.821)
  Cycle 17 Day 1 (n=85, 16) | 23.42 (4.603) | 22.25 (5.037)
  Cycle 17 Day 28 (n=80, 14) | 23.50 (4.424) | 21.75 (5.680)
  Cycle 18 Day 1 (n=79, 12) | 23.53 (4.428) | 21.71 (6.276)
  Cycle 18 Day 28 (n=70, 11) | 23.70 (4.410) | 21.27 (6.051)
  Cycle 19 Day 1 (n=71, 11) | 23.85 (4.270) | 21.30 (5.894)
  Cycle 19 Day 28 (n=61, 10) | 23.53 (4.641) | 20.73 (6.816)
  Cycle 20 Day 1 (n=63, 9) | 23.60 (4.045) | 21.26 (7.201)
  Cycle 20 Day 28 (n=52, 8) | 22.93 (4.898) | 20.67 (6.251)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Functional Assessment of Cancer Therapy-General (FACT-G) Social/Family Well Being (SWB) subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.214, 95% CI 2-sided [0.719 to 1.708]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.216, 95% CI 2-sided [0.729 to 1.703]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.217, 95% CI 2-sided [0.731 to 1.704]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.220, 95% CI 2-sided [0.730 to 1.710]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.221, 95% CI 2-sided [0.727 to 1.716]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.224, 95% CI 2-sided [0.716 to 1.732]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.225, 95% CI 2-sided [0.707 to 1.744]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.228, 95% CI 2-sided [0.687 to 1.769]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.229, 95% CI 2-sided [0.673 to 1.785]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.232, 95% CI 2-sided [0.646 to 1.818]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.233, 95% CI 2-sided [0.629 to 1.838]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 1.236, 95% CI 2-sided [0.595 to 1.876]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 1.237, 95% CI 2-sided [0.575 to 1.899]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 1.240, 95% CI 2-sided [0.537 to 1.942]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 1.241, 95% CI 2-sided [0.515 to 1.967]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 1.244, 95% CI 2-sided [0.474 to 2.013]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mean Difference (Final Values) = 1.245, 95% CI 2-sided [0.450 to 2.040]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; Mean Difference (Final Values) = 1.248, 95% CI 2-sided [0.406 to 2.089]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis; Mean Difference (Final Values) = 1.249, 95% CI 2-sided [0.382 to 2.116]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0074, Mixed Models Analysis; Mean Difference (Final Values) = 1.251, 95% CI 2-sided [0.336 to 2.167]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0092, Mixed Models Analysis; Mean Difference (Final Values) = 1.253, 95% CI 2-sided [0.310 to 2.196]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0132, Mixed Models Analysis; Mean Difference (Final Values) = 1.255, 95% CI 2-sided [0.262 to 2.248]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0159, Mixed Models Analysis; Mean Difference (Final Values) = 1.257, 95% CI 2-sided [0.236 to 2.278]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0213, Mixed Models Analysis; Mean Difference (Final Values) = 1.259, 95% CI 2-sided [0.187 to 2.332]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0248, Mixed Models Analysis; Mean Difference (Final Values) = 1.261, 95% CI 2-sided [0.160 to 2.362]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0318, Mixed Models Analysis; Mean Difference (Final Values) = 1.263, 95% CI 2-sided [0.110 to 2.416]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0360, Mixed Models Analysis; Mean Difference (Final Values) = 1.265, 95% CI 2-sided [0.083 to 2.447]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0443, Mixed Models Analysis; Mean Difference (Final Values) = 1.267, 95% CI 2-sided [0.032 to 2.502]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0493, Mixed Models Analysis; Mean Difference (Final Values) = 1.269, 95% CI 2-sided [0.004 to 2.533]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0587, Mixed Models Analysis; Mean Difference (Final Values) = 1.271, 95% CI 2-sided [-0.047 to 2.589]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0642, Mixed Models Analysis; Mean Difference (Final Values) = 1.273, 95% CI 2-sided [-0.075 to 2.620]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0746, Mixed Models Analysis; Mean Difference (Final Values) = 1.275, 95% CI 2-sided [-0.127 to 2.677]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0806, Mixed Models Analysis; Mean Difference (Final Values) = 1.276, 95% CI 2-sided [-0.155 to 2.708]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0917, Mixed Models Analysis; Mean Difference (Final Values) = 1.279, 95% CI 2-sided [-0.207 to 2.765]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0980, Mixed Models Analysis; Mean Difference (Final Values) = 1.280, 95% CI 2-sided [-0.236 to 2.797]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1095, Mixed Models Analysis; Mean Difference (Final Values) = 1.283, 95% CI 2-sided [-0.288 to 2.854]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1161, Mixed Models Analysis; Mean Difference (Final Values) = 1.284, 95% CI 2-sided [-0.318 to 2.886]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1280, Mixed Models Analysis; Mean Difference (Final Values) = 1.287, 95% CI 2-sided [-0.370 to 2.944]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1346, Mixed Models Analysis; Mean Difference (Final Values) = 1.288, 95% CI 2-sided [-0.399 to 2.976]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G SWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1466, Mixed Models Analysis; Mean Difference (Final Values) = 1.291, 95% CI 2-sided [-0.452 to 3.034]

15. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G): Emotional Well Being (EWB) Subscale
Description: Emotional well-being (EWB)subscale of the Functional Assessment of Cancer Therapy-General (FACT-G). Each question was answered on a five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Score = the sum score of the item scores in the subscale; range: 0 to 24; lower score indicates better emotional well-being.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (370, 352) | 17.15 (4.548) | 17.06 (4.609)
  Cycle 1 Day 28 (n=347, 318) | 17.76 (4.347) | 17.40 (5.123)
  Cycle 2 Day 1 (n=328, 249) | 18.46 (4.218) | 17.52 (4.560)
  Cycle 2 Day 28 (n=316, 237) | 18.46 (4.342) | 17.73 (4.637)
  Cycle 3 Day 1 (n=294, 200) | 18.82 (4.236) | 18.13 (4.603)
  Cycle 3 Day 28 (n=287, 196) | 18.53 (4.494) | 18.17 (4.704)
  Cycle 4 Day 1 (n=272, 152) | 19.04 (4.182) | 18.80 (4.246)
  Cycle 4 Day 28 (n=265, 142) | 18.76 (4.343) | 18.39 (4.378)
  Cycle 5 Day 1 (n=249, 120) | 19.18 (3.903) | 19.00 (4.062)
  Cycle 5 Day 28 (n=241, 109) | 18.63 (4.298) | 18.70 (4.144)
  Cycle 6 Day 1 (n=240, 99) | 18.99 (4.154) | 18.60 (4.338)
  Cycle 6 Day 28 (n=222, 99) | 18.73 (4.311) | 18.14 (4.747)
  Cycle 7 Day 1 (n=208, 77) | 19.08 (4.324) | 18.08 (5.010)
  Cycle 7 Day 28 (n=204, 75) | 18.69 (4.595) | 18.55 (4.691)
  Cycle 8 Day 1 (n=192, 67) | 19.33 (4.104) | 18.54 (4.613)
  Cycle 8 Day 28 (n=189, 62) | 18.98 (4.026) | 18.55 (4.734)
  Cycle 9 Day 1 (n=171, 51) | 19.25 (4.341) | 18.98 (4.654)
  Cycle 9 Day 28 (n=167, 46) | 18.93 (4.376) | 18.76 (4.831)
  Cycle 10 Day 1 (n=161, 50) | 19.32 (4.191) | 18.92 (4.548)
  Cycle 10 Day 28 (n=154, 45) | 18.71 (4.557) | 18.36 (4.778)
  Cycle 11 Day 1 (n=138, 35) | 18.92 (4.514) | 18.97 (4.225)
  Cycle 11 Day 28 (n=141, 33) | 19.10 (4.209) | 18.52 (5.316)
  Cycle 12 Day 1 (n=132, 30) | 19.14 (4.547) | 18.87 (4.547)
  Cycle 12 Day 28 (n=128, 31) | 19.06 (4.456) | 19.45 (4.178)
  Cycle 13 Day 1 (n=114, 27) | 19.38 (4.170) | 18.63 (4.853)
  Cycle 13 Day 28 (n=114, 27) | 19.39 (4.034) | 18.97 (3.993)
  Cycle 14 Day 1 (n=114, 26) | 19.55 (3.951) | 18.05 (4.814)
  Cycle 14 Day 28 (n=107, 25) | 19.23 (4.522) | 18.76 (4.085)
  Cycle 15 Day 1 (n=101, 21) | 19.57 (4.171) | 18.24 (4.795)
  Cycle 15 Day 28 (n=96, 20) | 19.41 (4.459) | 18.75 (4.447)
  Cycle 16 Day 1 (n=96, 19) | 19.54 (4.258) | 17.26 (5.675)
  Cycle 16 Day 28 (n=91, 18) | 19.33 (4.287) | 16.83 (5.113)
  Cycle 17 Day 1 (n=84, 17) | 19.95 (3.997) | 18.28 (5.151)
  Cycle 17 Day 28 (n=81, 14) | 19.66 (4.420) | 18.00 (5.218)
  Cycle 18 Day 1 (n=80, 12) | 19.64 (4.132) | 19.62 (4.971)
  Cycle 18 Day 28 (n=71, 11) | 19.34 (4.125) | 19.55 (4.677)
  Cycle 19 Day 1 (n=71, 11) | 19.94 (4.052) | 19.09 (5.224)
  Cycle 19 Day 28 (n=61, 10) | 19.61 (4.469) | 18.20 (6.630)
  Cycle 20 Day 1 (n=65, 9) | 20.00 (4.138) | 18.67 (5.788)
  Cycle 20 Day 28 (n=53, 9) | 19.75 (4.206) | 18.67 (6.384)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Functional Assessment of Cancer Therapy-General (FACT-G) Emotional Well Being (EWB) subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.929, 95% CI 2-sided [0.460 to 1.398]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.922, 95% CI [0.469 to 1.375]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.918, 95% CI [0.471 to 1.365]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.911, 95% CI [0.469 to 1.352]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.907, 95% CI [0.466 to 1.348]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.899, 95% CI [0.453 to 1.345]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.895, 95% CI [0.444 to 1.347]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 0.888, 95% CI [0.421 to 1.355]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 0.884, 95% CI [0.406 to 1.362]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 0.877, 95% CI [0.375 to 1.379]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = 0.873, 95% CI [0.356 to 1.390]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; Mean Difference (Final Values) = 0.866, 95% CI [0.318 to 1.414]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; Mean Difference (Final Values) = 0.862, 95% CI [0.295 to 1.428]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis; Mean Difference (Final Values) = 0.854, 95% CI [0.251 to 1.457]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis; Mean Difference (Final Values) = 0.850, 95% CI [0.226 to 1.475]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; Mean Difference (Final Values) = 0.843, 95% CI [0.179 to 1.508]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0168, Mixed Models Analysis; Mean Difference (Final Values) = 0.839, 95% CI [0.151 to 1.527]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0257, Mixed Models Analysis; Mean Difference (Final Values) = 0.832, 95% CI [0.101 to 1.563]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0318, Mixed Models Analysis; Mean Difference (Final Values) = 0.828, 95% CI [0.072 to 1.583]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0447, Mixed Models Analysis; Mean Difference (Final Values) = 0.821, 95% CI [0.019 to 1.622]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0529, Mixed Models Analysis; Mean Difference (Final Values) = 0.817, 95% CI [-0.010 to 1.643]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0696, Mixed Models Analysis; Mean Difference (Final Values) = 0.809, 95% CI [-0.065 to 1.683]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0797, Mixed Models Analysis; Mean Difference (Final Values) = 0.805, 95% CI [-0.095 to 1.706]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0994, Mixed Models Analysis; Mean Difference (Final Values) = 0.798, 95% CI [-0.151 to 1.747]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1110, Mixed Models Analysis; Mean Difference (Final Values) = 0.794, 95% CI [-0.182 to 1.770]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1328, Mixed Models Analysis; Mean Difference (Final Values) = 0.787, 95% CI [-0.239 to 1.813]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1454, Mixed Models Analysis; Mean Difference (Final Values) = 0.783, 95% CI [-0.271 to 1.836]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1686, Mixed Models Analysis; Mean Difference (Final Values) = 0.776, 95% CI [-0.329 to 1.880]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1817, Mixed Models Analysis; Mean Difference (Final Values) = 0.771, 95% CI [-0.361 to 1.904]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2055, Mixed Models Analysis; Mean Difference (Final Values) = 0.764, 95% CI [-0.419 to 1.948]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2188, Mixed Models Analysis; Mean Difference (Final Values) = 0.760, 95% CI [-0.452 to 1.972]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2427, Mixed Models Analysis; Mean Difference (Final Values) = 0.753, 95% CI [-0.510 to 2.016]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2559, Mixed Models Analysis; Mean Difference (Final Values) = 0.749, 95% CI [-0.543 to 2.041]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2794, Mixed Models Analysis; Mean Difference (Final Values) = 0.742, 95% CI [-0.602 to 2.086]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2923, Mixed Models Analysis; Mean Difference (Final Values) = 0.738, 95% CI [-0.635 to 2.111]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3152, Mixed Models Analysis; Mean Difference (Final Values) = 0.730, 95% CI [-0.695 to 2.156]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3276, Mixed Models Analysis; Mean Difference (Final Values) = 0.726, 95% CI [-0.728 to 2.181]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3497, Mixed Models Analysis; Mean Difference (Final Values) = 0.719, 95% CI [-0.788 to 2.227]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3616, Mixed Models Analysis; Mean Difference (Final Values) = 0.715, 95% CI [-0.822 to 2.252]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G EWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3827, Mixed Models Analysis; Mean Difference (Final Values) = 0.708, 95% CI [-0.882 to 2.298]

16. Secondary Outcome: Functional Assessment of Cancer Therapy-General (FACT-G): Functional Well Being (FWB) Subscale
Description: Functional well-being (FWB) subscale of the Functional Assessment of Cancer Therapy-General (FACT-G). Each question was answered on a five-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Score = the sum score of the item scores in the subscale; range: 0 to 28; higher score indicates greater functional well-being.
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=371, 353) | 18.93 (6.107) | 18.51 (6.389)
  Cycle 1 Day 28 (n=347, 318) | 17.92 (6.083) | 16.37 (6.694)
  Cycle 2 Day 1 (n=328, 249) | 18.78 (6.001) | 17.08 (6.279)
  Cycle 2 Day 28 (n=315, 238) | 18.37 (6.210) | 17.18 (6.673)
  Cycle 3 Day 1 (n=294, 200) | 19.51 (6.073) | 17.92 (6.251)
  Cycle 3 Day 28 (n=287, 195) | 18.58 (5.994) | 17.56 (6.762)
  Cycle 4 Day 1 (n=272, 152) | 19.93 (5.625) | 18.40 (6.382)
  Cycle 4 Day 28 (n=265, 142) | 18.86 (5.694) | 18.37 (6.430)
  Cycle 5 Day 1 (n=249, 120) | 20.27 (5.593) | 18.81 (5.697)
  Cycle 5 Day 28 (n=241, 109) | 19.02 (5.829) | 18.47 (6.065)
  Cycle 6 Day 1 (n=239, 99) | 19.74 (5.608) | 19.02 (6.114)
  Cycle 6 Day 28 (n=222, 99) | 19.21 (5.678) | 18.24 (6.273)
  Cycle 7 Day 1 (n=208, 79) | 19.69 (5.645) | 18.45 (6.761)
  Cycle 7 Day 28 (n=204, 75) | 19.12 (5.798) | 18.76 (6.036)
  Cycle 8 Day 1 (n=192, 67) | 20.29 (5.285) | 19.22 (5.828)
  Cycle 8 Day 28 (n=190, 62) | 19.33 (5.627) | 19.10 (6.098)
  Cycle 9 Day 1 (n=170, 51) | 19.87 (5.635) | 20.20 (5.455)
  Cycle 9 Day 28 (n=167, 46) | 19.27 (5.701) | 20.04 (5.929)
  Cycle 10 Day 1 (n=161, 50) | 19.95 (5.420) | 19.88 (5.903)
  Cycle 10 Day 28 (n=154, 46) | 19.22 (5.494) | 19.40 (6.126)
  Cycle 11 Day 1 (n=137, 35) | 19.81 (5.368) | 18.89 (6.014)
  Cycle 11 Day 28 (n=140, 33) | 19.12 (5.749) | 18.81 (6.441)
  Cycle 12 Day 1 (n=132, 30) | 19.98 (5.618) | 18.80 (6.599)
  Cycle 12 Day 28 (n=128, 31) | 19.42 (5.755) | 19.13 (6.270)
  Cycle 13 Day 1 (n=114, 27) | 20.02 (5.703) | 19.63 (6.918)
  Cycle 13 Day 28 (n=114, 27) | 19.65 (5.216) | 18.59 (6.795)
  Cycle 14 Day 1 (n=114, 26) | 20.04 (5.556) | 19.62 (6.020)
  Cycle 14 Day 28 (n=107, 25) | 19.07 (6.025) | 19.72 (6.662)
  Cycle 15 Day 1 (n=101, 21) | 20.13 (5.654) | 19.86 (6.327)
  Cycle 15 Day 28 (n=96, 20) | 19.24 (5.589) | 19.83 (5.736)
  Cycle 16 Day 1 (n=96, 19) | 19.80 (5.469) | 18.89 (6.154)
  Cycle 16 Day 28 (n=91, 18) | 19.53 (5.313) | 18.61 (6.464)
  Cycle 17 Day 1 (n=85, 17) | 20.20 (5.606) | 19.35 (6.103)
  Cycle 17 Day 28 (n=81, 14) | 19.67 (5.662) | 18.71 (6.557)
  Cycle 18 Day 1 (n=80, 12) | 19.76 (5.862) | 19.08 (7.317)
  Cycle 18 Day 28 (n=71, 11) | 19.47 (5.526) | 19.00 (7.155)
  Cycle 19 Day 1 (n=71, 11) | 20.18 (5.563) | 19.64 (7.500)
  Cycle 19 Day 28 (n=61, 10) | 19.59 (6.326) | 19.10 (8.048)
  Cycle 20 Day 1 (n=65, 9) | 20.50 (5.425) | 20.00 (7.826)
  Cycle 20 Day 28 (n=53, 9) | 20.15 (5.819) | 20.22 (7.694)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Functional Assessment of Cancer Therapy-General (FACT-G) Functional Well Being (FWB) subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.897, 95% CI 2-sided [1.261 to 2.533]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.924, 95% CI [1.309 to 2.539]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.939, 95% CI [1.331 to 2.546]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.965, 95% CI [1.363 to 2.568]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.980, 95% CI [1.376 to 2.584]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.007, 95% CI [1.392 to 2.622]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.022, 95% CI [1.396 to 2.647]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.048, 95% CI [1.397 to 2.700]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.063, 95% CI [1.394 to 2.732]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.090, 95% CI [1.383 to 2.797]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.105, 95% CI [1.374 to 2.836]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.132, 95% CI [1.353 to 2.910]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.146, 95% CI [1.339 to 2.954]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.173, 95% CI [1.311 to 3.036]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.188, 95% CI [1.294 to 3.082]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.215, 95% CI [1.260 to 3.169]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.230, 95% CI [1.241 to 3.219]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.256, 95% CI [1.203 to 3.309]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.271, 95% CI [1.182 to 3.361]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.298, 95% CI [1.142 to 3.454]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 2.313, 95% CI [1.119 to 3.507]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 2.340, 95% CI [1.076 to 3.603]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 2.354, 95% CI [1.052 to 3.657]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 2.381, 95% CI [1.008 to 3.754]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = 2.396, 95% CI [0.983 to 3.809]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Mean Difference (Final Values) = 2.423, 95% CI [0.938 to 3.908]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; Mean Difference (Final Values) = 2.438, 95% CI [0.912 to 3.963]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; Mean Difference (Final Values) = 2.464, 95% CI [0.866 to 4.063]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis; Mean Difference (Final Values) = 2.479, 95% CI [0.840 to 4.119]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0042, Mixed Models Analysis; Mean Difference (Final Values) = 2.506, 95% CI [0.792 to 4.219]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis; Mean Difference (Final Values) = 2.521, 95% CI [0.766 to 4.275]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; Mean Difference (Final Values) = 2.547, 95% CI [0.718 to 4.377]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; Mean Difference (Final Values) = 2.562, 95% CI [0.691 to 4.433]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; Mean Difference (Final Values) = 2.589, 95% CI [0.643 to 4.535]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0103, Mixed Models Analysis; Mean Difference (Final Values) = 2.604, 95% CI [0.616 to 4.592]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0125, Mixed Models Analysis; Mean Difference (Final Values) = 2.631, 95% CI [0.567 to 4.695]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0138, Mixed Models Analysis; Mean Difference (Final Values) = 2.645, 95% CI [0.539 to 4.752]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0164, Mixed Models Analysis; Mean Difference (Final Values) = 2.672, 95% CI [0.490 to 4.855]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0179, Mixed Models Analysis; Mean Difference (Final Values) = 2.687, 95% CI [0.462 to 4.912]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline FACT-G FWB subscale baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0208, Mixed Models Analysis; Mean Difference (Final Values) = 2.714, 95% CI [0.413 to 5.015]

17. Secondary Outcome: EuroQoL Five Dimension (EQ-5D) Health State Index
Description: EQ-5D Health State Index: a brief, self-administered generic health status instrument. Respondents were asked to describe their current health state on each of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety or depression) on a three-level scale (1=no problem, 2=some problem, and 3=extreme problem). A maximum score of 1 can be derived from these 5 dimensions by score conversion; range: -0.39 (worst health state)to 1.00 (best health state). This descriptive system classifies respondents into one of 243 possible distinct health states (EQ-5D descriptive system).
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=363, 352) | 0.76 (0.225) | 0.76 (0.234)
  Cycle 1 Day 28 (346, 315) | 0.72 (0.262) | 0.70 (0.274)
  Cycle 2 Day 1 (326, 244) | 0.78 (0.230) | 0.75 (0.231)
  Cycle 2 Day 28 (311, 233) | 0.73 (0.246) | 0.74 (0.230)
  Cycle 3 Day 1 (287, 200) | 0.78 (0.220) | 0.76 (0.222)
  Cycle 3 Day 28 (283, 195) | 0.75 (0.231) | 0.75 (0.218)
  Cycle 4 Day 1 (269, 150) | 0.80 (0.199) | 0.80 (0.190)
  Cycle 4 Day 28 (261, 142) | 0.76 (0.218) | 0.79 (0.216)
  Cycle 5 Day 1 (247, 120) | 0.80 (0.209) | 0.79 (0.194)
  Cycle 5 Day 28 (240, 106) | 0.76 (0.223) | 0.78 (0.201)
  Cycle 6 Day 1 (240, 98) | 0.80 (0.249) | 0.80 (0.178)
  Cycle 6 Day 28 (224, 100) | 0.77 (0.206) | 0.80 (0.187)
  Cycle 7 Day 1 (205, 79) | 0.81 (0.192) | 0.80 (0.185)
  Cycle 7 Day 28 (204, 74) | 0.77 (0.221) | 0.81 (0.156)
  Cycle 8 Day 1 (192, 68) | 0.82 (0.180) | 0.82 (0.158)
  Cycle 8 Day 28 (190, 61) | 0.77 (0.222) | 0.81 (0.163)
  Cycle 9 Day 1 (170, 51) | 0.80 (0.196) | 0.84 (0.162)
  Cycle 9 Day 28 (168, 45) | 0.78 (0.194) | 0.84 (0.147)
  Cycle 10 Day 1 (161, 50) | 0.81 (0.209) | 0.85 (0.161)
  Cycle 10 Day 28 (153, 46) | 0.78 (0.200) | 0.82 (0.185)
  Cycle 11 Day 1 (138, 34) | 0.80 (0.192) | 0.85 (0.159)
  Cycle 11 Day 28 (138, 32) | 0.75 (0.189) | 0.84 (0.185)
  Cycle 12 Day 1 (132, 31) | 0.81 (0.187) | 0.82 (0.283)
  Cycle 12 Day 28 (127, 31) | 0.77 (0.182) | 0.85 (0.165)
  Cycle 13 Day 1 (114, 26) | 0.81 (0.176) | 0.83 (0.231)
  Cycle 13 Day 28 (115, 27) | 0.77 (0.186) | 0.82 (0.260)
  Cycle 14 Day 1 (114, 25) | 0.81 (0.181) | 0.86 (0.148)
  Cycle 14 Day 28 (107, 24) | 0.75 (0.224) | 0.87 (0.160)
  Cycle 15 Day 1 (100, 21) | 0.80 (0.190) | 0.88 (0.146)
  Cycle 15 Day 28 (95, 20) | 0.75 (0.209) | 0.88 (0.141)
  Cycle 16 Day 1 (96, 19) | 0.79 (0.194) | 0.84 (0.163)
  Cycle 16 Day 28 (93, 18) | 0.76 (0.181) | 0.83 (0.164)
  Cycle 17 Day 1 (84, 15) | 0.79 (0.194) | 0.88 (0.169)
  Cycle 17 Day 28 (82, 14) | 0.77 (0.168) | 0.83 (0.174)
  Cycle 18 Day 1 (80, 12) | 0.81 (0.187) | 0.86 (0.274)
  Cycle 18 Day 28 (71, 10) | 0.76 (0.166) | 0.84 (0.279)
  Cycle 19 Day 1 (69, 11) | 0.81 (0.183) | 0.88 (0.184)
  Cycle 19 Day 28 (62, 11) | 0.78 (0.165) | 0.72 (0.436)
  Cycle 20 Day 1 (63, 8) | 0.81 (0.162) | 0.85 (0.182)
  Cycle 20 Day 28 (54, 9) | 0.77 (0.181) | 0.86 (0.215)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EuroQoL Five Dimension (EQ-5D): Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [0.022 to 0.076]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 0.048, 95% CI [0.022 to 0.075]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 0.048, 95% CI [0.022 to 0.074]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 0.047, 95% CI [0.021 to 0.072]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 0.046, 95% CI [0.021 to 0.072]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI [0.020 to 0.071]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI [0.019 to 0.070]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 95% CI [0.017 to 0.070]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = 0.043, 95% CI [0.016 to 0.070]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI [0.014 to 0.070]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI [0.013 to 0.070]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI [0.011 to 0.071]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0105, Mixed Models Analysis; Mean Difference (Final Values) = 0.040, 95% CI [0.009 to 0.071]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0179, Mixed Models Analysis; Mean Difference (Final Values) = 0.039, 95% CI [0.007 to 0.072]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0236, Mixed Models Analysis; Mean Difference (Final Values) = 0.039, 95% CI [0.005 to 0.072]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0370, Mixed Models Analysis; Mean Difference (Final Values) = 0.038, 95% CI [0.002 to 0.073]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0464, Mixed Models Analysis; Mean Difference (Final Values) = 0.037, 95% CI [0.001 to 0.074]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0667, Mixed Models Analysis; Mean Difference (Final Values) = 0.036, 95% CI [-0.002 to 0.075]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0800, Mixed Models Analysis; Mean Difference (Final Values) = 0.036, 95% CI [-0.004 to 0.076]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1070, Mixed Models Analysis; Mean Difference (Final Values) = 0.035, 95% CI [-0.007 to 0.077]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1237, Mixed Models Analysis; Mean Difference (Final Values) = 0.034, 95% CI [-0.009 to 0.078]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1561, Mixed Models Analysis; Mean Difference (Final Values) = 0.033, 95% CI [-0.013 to 0.079]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.1752, Mixed Models Analysis; Mean Difference (Final Values) = 0.033, 95% CI [-0.015 to 0.080]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2112, Mixed Models Analysis; Mean Difference (Final Values) = 0.032, 95% CI [-0.018 to 0.081]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2319, Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI [-0.020 to 0.082]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2698, Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI [-0.023 to 0.084]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.2910, Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI [-0.025 to 0.085]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3293, Mixed Models Analysis; Mean Difference (Final Values) = 0.029, 95% CI [-0.029 to 0.086]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3504, Mixed Models Analysis; Mean Difference (Final Values) = 0.028, 95% CI [-0.031 to 0.087]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.3881, Mixed Models Analysis; Mean Difference (Final Values) = 0.027, 95% CI [-0.034 to 0.089]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.4086, Mixed Models Analysis; Mean Difference (Final Values) = 0.027, 95% CI [-0.036 to 0.090]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.4449, Mixed Models Analysis; Mean Difference (Final Values) = 0.026, 95% CI [-0.040 to 0.091]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.4646, Mixed Models Analysis; Mean Difference (Final Values) = 0.025, 95% CI [-0.042 to 0.092]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.4990, Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI [-0.046 to 0.094]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.5176, Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI [-0.048 to 0.095]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.5501, Mixed Models Analysis; Mean Difference (Final Values) = 0.023, 95% CI [-0.051 to 0.097]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.5675, Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI [-0.054 to 0.098]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.5979, Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI [-0.057 to 0.099]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.6141, Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI [-0.059 to 0.100]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-5D Health state index baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.6424, Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 95% CI [-0.063 to 0.102]

18. Secondary Outcome: Euro-QoL Visual Analog Scale (EQ-VAS)
Description: EQ-VAS: overall self-rating rating of the patient's current health state using a 20 cm Visual Analog Scale (EQ-VAS), also called the health state thermometer) is a metric measurement (in 2 mm interval) from the visual analog scale which ranges between 0 (worse imaginable health state) and 100 (best imaginable health state).
Time Frame: Day 1 & 28 of each cycle: duration of treatment phase
Population: ITT; N=number of subjects with evaluable data; n=number of subjects with evaluable data at observation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
scores on scale
  Baseline (n=365, 352) | 73.80 (18.498) | 71.43 (19.507)
  Cycle 1 Day 28 (n=347, 315) | 69.35 (18.992) | 67.66 (20.058)
  Cycle 2 Day 1 (n=323, 247) | 75.05 (17.964) | 70.45 (17.653)
  Cycle 2 Day 28 (n=314, 237) | 72.06 (18.297) | 70.70 (18.271)
  Cycle 3 Day 1 (n=293, 198) | 76.23 (17.171) | 72.68 (17.162)
  Cycle 3 Day 28 (n=287, 193) | 72.33 (18.472) | 71.45 (18.315)
  Cycle 4 Day 1 (n=270, 152) | 77.46 (16.024) | 72.74 (17.678)
  Cycle 4 Day 28 (n=264, 139) | 75.15 (16.406) | 72.20 (18.098)
  Cycle 5 Day 1 (n=248, 118) | 79.83 (13.554) | 73.44 (16.204)
  Cycle 5 Day 28 (n=240, 104) | 75.13 (16.771) | 72.57 (16.007)
  Cycle 6 Day 1 (n=237, 99) | 78.83 (15.359) | 73.68 (16.537)
  Cycle 6 Day 28 (n=223, 98) | 76.81 (15.204) | 72.26 (18.452)
  Cycle 7 Day 1 (n=209, 77) | 79.39 (14.601) | 73.80 (18.868)
  Cycle 7 Day 28 (n=201, 74) | 76.09 (16.693) | 73.46 (17.380)
  Cycle 8 Day 1 (n=192, 67) | 81.34 (13.020) | 74.27 (18.067)
  Cycle 8 Day 28 (n=191, 60) | 77.53 (14.374) | 74.33 (18.407)
  Cycle 9 Day 1 (n=172, 50) | 80.08 (13.812) | 77.66 (15.987)
  Cycle 9 Day 28 (n=168, 46) | 76.24 (15.740) | 76.57 (17.924)
  Cycle 10 Day 1 (n=160, 50) | 79.18 (14.912) | 76.64 (17.886)
  Cycle 10 Day 28 (n=154, 45) | 76.44 (16.106) | 76.69 (19.123)
  Cycle 11 Day 1 (n=138, 34) | 79.72 (15.685) | 75.06 (20.179)
  Cycle 11 Day 28 (n=141, 33) | 76.81 (15.128) | 72.21 (23.202)
  Cycle 12 Day 1 (n=130, 31) | 80.84 (14.150) | 75.19 (22.020)
  Cycle 12 Day 28 (n=128, 31) | 76.71 (14.986) | 73.84 (20.775)
  Cycle 13 Day 1 (n=114, 27) | 80.59 (14.875) | 77.52 (17.738)
  Cycle 13 Day 28 (n=115, 27) | 77.22 (14.715) | 73.56 (23.523)
  Cycle 14 Day 1 (n=114, 26) | 80.39 (14.477) | 76.69 (16.601)
  Cycle 14 Day 28 (n=107, 25) | 76.53 (15.933) | 76.44 (18.890)
  Cycle 15 Day 1 (n=101, 21) | 80.50 (14.361) | 76.62 (19.075)
  Cycle 15 Day 28 (n=96, 20) | 76.51 (15.141) | 76.50 (18.841)
  Cycle 16 Day 1 (n=96, 19) | 79.85 (15.632) | 74.84 (21.680)
  Cycle 16 Day 28 (n=92, 18) | 75.51 (17.687) | 73.11 (21.202)
  Cycle 17 Day 1 (n=84, 17) | 80.74 (15.706) | 76.94 (21.256)
  Cycle 17 Day 28 (n=82, 14) | 77.10 (16.612) | 72.86 (22.593)
  Cycle 18 Day 1 (n=78, 12) | 80.40 (14.658) | 74.42 (25.065)
  Cycle 18 Day 28 (n=70, 11) | 77.76 (16.142) | 73.82 (24.140)
  Cycle 19 Day 1 (n=70, 11) | 81.47 (15.330) | 79.27 (20.283)
  Cycle 19 Day 28 (n=62, 11) | 77.05 (18.676) | 68.55 (29.717)
  Cycle 20 Day 1 (n=65, 9) | 81.10 (15.404) | 76.00 (21.494)
  Cycle 20 Day 28 (n=54, 9) | 76.85 (16.863) | 75.44 (25.060)
Statistical Analysis 1: Comparison: SU011248 vs IFN-α; Cycle 1 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline Euro-QoL Visual Analog Scale (EQ-VAS) baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.026, 95% CI 2-sided [2.088 to 5.965]
Statistical Analysis 2: Comparison: SU011248 vs IFN-α; Cycle 1 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.165, 95% CI [2.269 to 6.061]
Statistical Analysis 3: Comparison: SU011248 vs IFN-α; Cycle 2 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.243, 95% CI [2.358 to 6.128]
Statistical Analysis 4: Comparison: SU011248 vs IFN-α; Cycle 2 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.382, 95% CI [2.494 to 6.269]
Statistical Analysis 5: Comparison: SU011248 vs IFN-α; Cycle 3 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.459, 95% CI [2.558 to 6.361]
Statistical Analysis 6: Comparison: SU011248 vs IFN-α; Cycle 3 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.598, 95% CI [2.650 to 6.547]
Statistical Analysis 7: Comparison: SU011248 vs IFN-α; Cycle 4 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.676, 95% CI [2.689 to 6.662]
Statistical Analysis 8: Comparison: SU011248 vs IFN-α; Cycle 4 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.815, 95% CI [2.741 to 6.889]
Statistical Analysis 9: Comparison: SU011248 vs IFN-α; Cycle 5 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.892, 95% CI [2.760 to 7.024]
Statistical Analysis 10: Comparison: SU011248 vs IFN-α; Cycle 5 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.031, 95% CI [2.780 to 7.283]
Statistical Analysis 11: Comparison: SU011248 vs IFN-α; Cycle 6 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.109, 95% CI [2.783 to 7.435]
Statistical Analysis 12: Comparison: SU011248 vs IFN-α; Cycle 6 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.248, 95% CI [2.776 to 7.720]
Statistical Analysis 13: Comparison: SU011248 vs IFN-α; Cycle 7 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.325, 95% CI [2.767 to 7.884]
Statistical Analysis 14: Comparison: SU011248 vs IFN-α; Cycle 7 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.464, 95% CI [2.741 to 8.188]
Statistical Analysis 15: Comparison: SU011248 vs IFN-α; Cycle 8 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.542, 95% CI [2.723 to 8.361]
Statistical Analysis 16: Comparison: SU011248 vs IFN-α; Cycle 8 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 5.681, 95% CI [2.683 to 8.679]
Statistical Analysis 17: Comparison: SU011248 vs IFN-α; Cycle 9 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 5.758, 95% CI [2.657 to 8.859]
Statistical Analysis 18: Comparison: SU011248 vs IFN-α; Cycle 9 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 5.898, 95% CI [2.607 to 9.188]
Statistical Analysis 19: Comparison: SU011248 vs IFN-α; Cycle 10 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 5.975, 95% CI [2.576 to 9.374]
Statistical Analysis 20: Comparison: SU011248 vs IFN-α; Cycle 10 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = 6.114, 95% CI [2.517 to 9.711]
Statistical Analysis 21: Comparison: SU011248 vs IFN-α; Cycle 11 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = 6.191, 95% CI [2.482 to 9.900]
Statistical Analysis 22: Comparison: SU011248 vs IFN-α; Cycle 11 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 6.331, 95% CI [2.417 to 10.244]
Statistical Analysis 23: Comparison: SU011248 vs IFN-α; Cycle 12 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 6.408, 95% CI [2.379 to 10.436]
Statistical Analysis 24: Comparison: SU011248 vs IFN-α; Cycle 12 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; Mean Difference (Final Values) = 6.547, 95% CI [2.309 to 10.785]
Statistical Analysis 25: Comparison: SU011248 vs IFN-α; Cycle 13 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; Mean Difference (Final Values) = 6.624, 95% CI [2.269 to 10.980]
Statistical Analysis 26: Comparison: SU011248 vs IFN-α; Cycle 13 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; Mean Difference (Final Values) = 6.764, 95% CI [2.195 to 11.332]
Statistical Analysis 27: Comparison: SU011248 vs IFN-α; Cycle 14 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0042, Mixed Models Analysis; Mean Difference (Final Values) = 6.841, 95% CI [2.153 to 11.529]
Statistical Analysis 28: Comparison: SU011248 vs IFN-α; Cycle 14 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis; Mean Difference (Final Values) = 6.980, 95% CI [2.076 to 11.884]
Statistical Analysis 29: Comparison: SU011248 vs IFN-α; Cycle 15 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; Mean Difference (Final Values) = 7.057, 95% CI [2.032 to 12.083]
Statistical Analysis 30: Comparison: SU011248 vs IFN-α; Cycle 15 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0072, Mixed Models Analysis; Mean Difference (Final Values) = 7.197, 95% CI [1.953 to 12.441]
Statistical Analysis 31: Comparison: SU011248 vs IFN-α; Cycle 16 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0079, Mixed Models Analysis; Mean Difference (Final Values) = 7.274, 95% CI [1.908 to 12.640]
Statistical Analysis 32: Comparison: SU011248 vs IFN-α; Cycle 16 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Mean Difference (Final Values) = 7.413, 95% CI [1.826 to 13.000]
Statistical Analysis 33: Comparison: SU011248 vs IFN-α; Cycle 17 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis; Mean Difference (Final Values) = 7.491, 95% CI [1.780 to 13.201]
Statistical Analysis 34: Comparison: SU011248 vs IFN-α; Cycle 17 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis; Mean Difference (Final Values) = 7.630, 95% CI [1.697 to 13.562]
Statistical Analysis 35: Comparison: SU011248 vs IFN-α; Cycle 18 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0126, Mixed Models Analysis; Mean Difference (Final Values) = 7.707, 95% CI [1.650 to 13.764]
Statistical Analysis 36: Comparison: SU011248 vs IFN-α; Cycle 18 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0144, Mixed Models Analysis; Mean Difference (Final Values) = 7.846, 95% CI [1.565 to 14.127]
Statistical Analysis 37: Comparison: SU011248 vs IFN-α; Cycle 19 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0153, Mixed Models Analysis; Mean Difference (Final Values) = 7.924, 95% CI [1.518 to 14.329]
Statistical Analysis 38: Comparison: SU011248 vs IFN-α; Cycle 19 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0172, Mixed Models Analysis; Mean Difference (Final Values) = 8.063, 95% CI [1.432 to 14.693]
Statistical Analysis 39: Comparison: SU011248 vs IFN-α; Cycle 20 Day 1: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0182, Mixed Models Analysis; Mean Difference (Final Values) = 8.140, 95% CI [1.384 to 14.896]
Statistical Analysis 40: Comparison: SU011248 vs IFN-α; Cycle 20 Day 28: Differences in effect estimates between treatment arms. Repeated measures mixed-effects model with an intercept term, treatment, time since randomization, treatment-by-time interaction, and baseline EQ-VAS baseline score (intercept and time since randomization are included as random effects); Test type: Superiority or Other; p = 0.0201, Mixed Models Analysis; Mean Difference (Final Values) = 8.279, 95% CI [1.297 to 15.261]

19. Secondary Outcome: Plasma Concentrations of Soluble Proteins: Plasma VEGF-A, Plasma VEGF-C, Plasma sVEGFR-3, PLASMA IL-8, and PLASMA bFGF That May be Associated With Tumor Proliferation or Angiogenesis
Description: Plasma concentrations of soluble proteins that may be associated with tumor proliferation or angiogenesis collected from a subset of patients were analyzed by enzyme-linked immunosorbent assay (ELISA) analysis. Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio = plasma concentration of soluble protein (picograms per milliliter [pg/ml]) at timepoint / concentration of soluble protein (pg/ml) at baseline. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Day 1 & Day 28, Cycle 1 to Cycle 4
Population: Pharmacodynamic analyses performed at selected sites on AT population who had at least one pharmacokinetic sample; n= SU011248, INF-α; Abbreviations: C: Cycle, D: Day, VEGF: vascular endothelial growth factor, sVEGFR-3: soluble vascular endothelial growth factor Receptor-3, IL-8: interleukin-8, bFGF: basic fibroblast growth factor.
  .
Measure: Mean (Standard Deviation); unit: pg/ml and ratio to Baseline
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 35 | 31
pg/ml and ratio to Baseline
  Plasma VEGF-A: Baseline (n=33, 31) | 101.9 (184.3) | 109.0 (242.4)
  Plasma VEGF-A: C1D28: C1D1 (n=31, 26) | 4.280 (2.619) | 1.134 (0.683)
  Plasma VEGF-A: C2D1: C1D1 (n=32, 21) | 1.161 (0.624) | 1.171 (0.527)
  Plasma VEGF-A: C2D28: C1D1 (n=31, 20) | 5.851 (4.345) | 1.153 (0.517)
  Plasma VEGF-A: C3D1: C1D1 (n=27, 15) | 1.630 (1.685) | 1.253 (0.483)
  Plasma VEGF-A: C3D28: C1D1 (n=28, 15) | 5.236 (3.333) | 1.149 (0.570)
  Plasma VEGF-A: C4D1: C1D1 (n=27, 12) | 1.486 (1.125) | 1.209 (0.654)
  Plasma VEGF-A: C4D28: C1D1 (n=25, 11) | 4.924 (3.679) | 1.008 (0.372)
  Plasma VEGF-C: Baseline (n=35, 31) | 556.4 (311.7) | 651.2 (552.3)
  Plasma VEGF-C: C1D28: C1D1 (n=31, 26) | 0.945 (0.428) | 1.165 (0.606)
  Plasma VEGF-C: C2D1:C1D1 (n=30, 21) | 1.045 (0.623) | 1.177 (0.464)
  Plasma VEGF-C: C2D28:C1D1 (n=31, 19) | 0.871 (0.511) | 1.081 (0.410)
  Plasma VEGF-C: C3D1:C1D1 (n=28, 15) | 1.159 (0.659) | 1.174 (0.588)
  Plasma VEGF-C: C3D28:C1D1 (n=28, 15) | 1.043 (0.926) | 1.054 (0.586)
  Plasma VEGF-C: C4D1:C1D1 (n=28, 12) | 1.243 (1.304) | 1.382 (0.799)
  Plasma VEGF-C: C4:D28:C1D1 (n=26, 11) | 1.207 (1.269) | 1.139 (0.403)
  PLASMA sVEGFR-3: Baseline (n=29, 30) | 44049.3 (20168.2) | 40317.7 (12938.3)
  PLASMA sVEGFR-3: C1D28:C1D1 (n=27, 25) | 0.473 (0.185) | 1.068 (0.292)
  PLASMA sVEGFR-3: C2D1:C1D1 (n=28, 20) | 0.787 (0.172) | 1.075 (0.331)
  PLASMA sVEGFR-3: C2D28:C1D1 (n=28, 19) | 0.407 (0.173) | 1.150 (0.355)
  PLASMA sVEGFR-3: C3D1:C1D1 (n=25, 14) | 0.800 (0.309) | 1.015 (0.210)
  PLASMA sVEGFR-3: C3D28:C1D1 (n=25, 14) | 0.427 (0.194) | 1.042 (0.349)
  PLASMA sVEGFR-3: C4D1:C1D1 (n=24, 11) | 0.846 (0.380) | 1.183 (0.333)
  PLASMA sVEGFR-3: C4:D28:C1D1 (n=23, 10) | 0.486 (0.265) | 1.044 (0.141)
  PLASMA IL-8: Baseline (n=31, 29) | 10.1 (9.7) | 18.6 (32.0)
  PLASMA IL-8: C1D28:C1D1 (n=29, 25) | 2.815 (1.340) | 2.297 (2.036)
  PLASMA IL-8: C2D1:C1D1 (n=29, 20) | 1.716 (0.630) | 1.579 (0.688)
  PLASMA IL-8: C2D28:C1D1 (n=29, 19) | 2.423 (1.514) | 1.858 (0.849)
  PLASMA IL-8: C3D1:C1D1 (n=26, 15) | 2.788 (2.781) | 1.531 (0.693)
  PLASMA IL-8: C3D28:C1D1 (n=26, 14) | 2.574 (1.726) | 1.999 (0.964)
  PLASMA IL-8: C4D1:C1D1 (n=26, 12) | 1.934 (1.372) | 1.662 (0.736)
  PLASMA IL-8: C4:D28:C1D1 (n=25, 11) | 2.549 (1.489) | 2.492 (2.023)
  PLASMA bFGF: Baseline (n=21, 2) | 13.1 (13.1) | 13.6 (16.8)
  PLASMA bFGF: C1D28:C1D1 (n=15, 1) | 2.762 (5.087) | 0.429 (0)
  PLASMA bFGF: C2D1:C1D1 (n=13, 1) | 1.370 (1.800) | 0.157 (0)

20. Secondary Outcome: Plasma Concentrations of Soluble Proteins: Plasma Basic Fibroblast Growth Factor (bFGF) That May be Associated With Tumor Proliferation or Angiogenesis
Description: as for outcome 19
Time Frame: Day 1 & Day 28, Cycle 1 to Cycle 4
Population: Pharmacodynamic analyses performed at selected sites on AT population who had at least one PK (pharmacokinetic) sample; n = subjects with evaluable data at observation, SU011248 and INF-α treatment groups, respectively. Abbreviations: C = Cycle, D = Day, bFGF: basic fibroblast growth factor.
Measure: Mean (Standard Deviation); unit: pg/ml and ratio to Baseline
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 14 | 0
pg/ml and ratio to Baseline
  PLASMA bFGF: C2D28:C1D1 (n=14, 0) | 0.760 (0.604) |
  PLASMA bFGF: C3D1:C1D1 (n=12, 0) | 1.582 (2.622) |
  PLASMA bFGF: C3D28:C1D1 (n=12, 0) | 1.671 (2.109) |
  PLASMA bFGF: C4D1:C1D1 (n=14, 0) | 2.895 (4.252) |
  PLASMA bFGF: C4:D28:C1D1 (n=10, 0) | 0.803 (0.799) |

21. Secondary Outcome: Incremental Cost Effectiveness Ratio (ICER)
Description: Incremental cost effectiveness ratio (ICER) of sunitinib compared to IFN-a as first-line treatment for MRCC, defined as the ratio of the incremental cost of treatment over the incremental effectiveness; effectiveness measured as quality adjusted life year (QALY) gain. This objective was not addressed in the clinical study report, but an interim analysis of cost-effectiveness was presented separately. These results were not available for inclusion at the time of this posting.
Time Frame: post study measurement
Measure: Number; unit: ratio
Arm/Group | SU011248 | IFN-α
Number analyzed (Participants) | 375 | 375
ratio | 0 | 0

22. Secondary Outcome: Ctrough Concentrations of SU011248
Description: Subject observed Ctrough (trough drug) concentrations of SU011248 per cycle and study day determined by plasma trough samples collected from a subset of patients. Steady-state observed trough concentrations were dose corrected to the starting dose (reference dose) where appropriate. Concentrations below the limits of quantitation (BLQ) were set to 0. Ctrough = minimum (trough) plasma concentration (nanograms per milliliter [ng/mL]).
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: As treated (AT) population: all patients who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received. Pharmacokinetic (PK) analyses were performed on the AT population who had at least one PK sample. n=number of subjects with evaluable trough samples.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- SU011248: 50 mg taken orally once a day for 4 weeks followed by a 2-week off treatment cycle. Intra-subject dose reduction to 35.5 mg/day and 25 mg/day was allowed depending on type and severity of toxicity encountered.
Arm/Group | SU011248
Number analyzed (Participants) | 45
ng/mL
  Cycle 1, Day 28 (n=31) | 57.26 (31.37)
  Cycle 2, Day 28 (n=36) | 57.59 (28.59)
  Cycle 3, Day 28 (n=36) | 50.26 (24.89)
  Cycle 4, Day 28 (n=32) | 45.05 (23.76)
  Dose-Corrected: Cycle 1, Day 28 (n=24) | 64.22 (31.40)
  Dose-Corrected: Cycle 2, Day 28 (n=28) | 59.90 (26.42)
  Dose-Corrected: Cycle 3, Day 28 (n=27) | 58.45 (29.39)
  Dose-Corrected: Cycle 4, Day 28 (n=26) | 54.31 (30.70)

23. Secondary Outcome: Ctrough Concentrations of Metabolite SU012662
Description: Subject observed Ctrough (trough drug) concentrations of active metabolite SU012662 per cycle and study day determined by plasma trough samples collected from a subset of patients. Steady-state observed trough concentrations were dose corrected to the starting dose (reference dose) where appropriate. Concentrations below the limits of quantitation (BLQ) were set to 0. Ctrough = minimum (trough) plasma concentration (nanograms per milliliter [ng/mL]).
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- SU012662: Active metabolite of SU011248
Arm/Group | SU012662
Number analyzed (Participants) | 45
ng/mL
  Cycle 1, Day 28 (n=31) | 27.10 (17.28)
  Cycle 2, Day 28 (n=36) | 27.35 (15.42)
  Cycle 3, Day 28 (n=36) | 26.11 (16.15)
  Cycle 4, Day 28 (n=32) | 22.11 (12.67)
  Dose-Corrected: Cycle 1, Day 28 (n=24) | 28.21 (19.01)
  Dose-Corrected: Cycle 2, Day 28 (n=28) | 28.32 (13.74)
  Dose-Corrected: Cycle 3, Day 28 (n=27) | 29.04 (19.07)
  Dose-Corrected: Cycle 4, Day 28 (n=26) | 25.99 (16.25)

24. Secondary Outcome: Ctrough Concentrations of SU011248 and Active Metabolite SU012662
Description: Subject observed Ctrough (trough drug) concentrations of total drug (SU011248 and its active metabolite SU012662) per cycle and study day determined by plasma trough samples collected from a subset of patients. Steady-state observed trough concentrations were dose corrected to the starting dose (reference dose) where appropriate. Concentrations below the limits of quantitation (BLQ) were set to 0. Ctrough = minimum (trough) plasma concentration (nanograms per milliliter [ng/mL]).
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: As treated (AT) population: all patients who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received. Pharmacokinetic (PK) analyses were performed on the AT population who had at least one PK sample. n=number of subjects with evaluable trough samples at observation.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Total Drug: SU011248 and SU012662: SU011248 and active metabolite SU012662
Arm/Group | Total Drug: SU011248 and SU012662
Number analyzed (Participants) | 45
ng/mL
  Cycle 1, Day 28 (n=31) | 84.36 (46.06)
  Cycle 2, Day 28 (n=36) | 84.94 (41.18)
  Cycle 3, Day 28 (n=36) | 76.37 (38.86)
  Cycle 4, Day 28 (n=32) | 67.15 (34.13)
  Dose-Corrected: Cycle 1, Day 28 (n=24) | 92.43 (48.08)
  Dose-Corrected: Cycle 2, Day 28 (n=28) | 88.22 (36.34)
  Dose-Corrected: Cycle 3, Day 28 (n=27) | 87.49 (45.85)
  Dose-Corrected: Cycle 4, Day 28 (n=27) | 80.30 (44.76)

ADVERSE EVENTS:
Arm/Group | SU011248 | IFN-α
Serious Adverse Events (participants affected / at risk) | 170/375 | 93/360
Other Adverse Events (participants affected / at risk) | 368/375 | 344/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU011248 (N=375) | IFN-α (N=360)
Anaemia (Blood and lymphatic system disorders) | 14 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 8 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 17 | 15
Asthenia (General disorders) | 16 | 5
Chest pain (General disorders) | 7 | 6
General physical health deterioration (General disorders) | 5 | 0
Pyrexia (General disorders) | 5 | 0
Condition aggravated (General disorders) | 3 | 2
Fatigue (General disorders) | 3 | 5
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 2
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Ejection fraction decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 11 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 3 | 1
Spinal cord compression (Nervous system disorders) | 3 | 1
Epilepsy (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Monoparesis (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Incoherent (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Mental status changes (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Bone graft (Surgical and medical procedures) | 1 | 0
Hepatectomy (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Pleurectomy (Surgical and medical procedures) | 1 | 0
Vertebroplasty (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 8 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SU011248 (N=375) | IFN-α (N=360)
Anaemia (Blood and lymphatic system disorders) | 75 | 55
Leukopenia (Blood and lymphatic system disorders) | 40 | 16
Lymphopenia (Blood and lymphatic system disorders) | 19 | 21
Neutropenia (Blood and lymphatic system disorders) | 69 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 69 | 15
Hypothyroidism (Endocrine disorders) | 57 | 3
Abdominal pain (Gastrointestinal disorders) | 64 | 28
Abdominal pain upper (Gastrointestinal disorders) | 52 | 10
Constipation (Gastrointestinal disorders) | 85 | 48
Diarrhoea (Gastrointestinal disorders) | 245 | 76
Dry mouth (Gastrointestinal disorders) | 50 | 27
Dyspepsia (Gastrointestinal disorders) | 128 | 16
Flatulence (Gastrointestinal disorders) | 52 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 47 | 3
Glossodynia (Gastrointestinal disorders) | 39 | 2
Haemorrhoids (Gastrointestinal disorders) | 38 | 6
Nausea (Gastrointestinal disorders) | 215 | 146
Oral pain (Gastrointestinal disorders) | 54 | 2
Stomatitis (Gastrointestinal disorders) | 113 | 12
Stomatitis (Gastrointestinal disorders) | 144 | 60
Asthenia (General disorders) | 91 | 79
Chest pain (General disorders) | 45 | 21
Chills (General disorders) | 52 | 111
Fatigue (General disorders) | 230 | 200
Influenza like illness (General disorders) | 18 | 54
Mucosal inflammation (General disorders) | 100 | 7
Oedema peripheral (General disorders) | 90 | 17
Pain (General disorders) | 35 | 20
Pyrexia (General disorders) | 80 | 134
Nasopharyngitis (Infections and infestations) | 54 | 8
Upper respiratory tract infection (Infections and infestations) | 42 | 9
Ejection fraction decreased (Investigations) | 60 | 19
Weight decreased (Investigations) | 60 | 59
Anorexia (Metabolism and nutrition disorders) | 154 | 112
Decreased appetite (Metabolism and nutrition disorders) | 44 | 44
Dehydration (Metabolism and nutrition disorders) | 27 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 110 | 68
Back pain (Musculoskeletal and connective tissue disorders) | 103 | 52
Bone pain (Musculoskeletal and connective tissue disorders) | 27 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 28 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 50 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 46 | 68
Pain in extremity (Musculoskeletal and connective tissue disorders) | 100 | 30
Dizziness (Nervous system disorders) | 43 | 50
Dysgeusia (Nervous system disorders) | 174 | 53
Headache (Nervous system disorders) | 86 | 69
Paraesthesia (Nervous system disorders) | 35 | 7
Anxiety (Psychiatric disorders) | 24 | 18
Depression (Psychiatric disorders) | 40 | 51
Insomnia (Psychiatric disorders) | 56 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 50
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 95 | 67
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 79 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 51 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 51 | 34
Dry skin (Skin and subcutaneous tissue disorders) | 85 | 26
Erythema (Skin and subcutaneous tissue disorders) | 46 | 5
Hair colour changes (Skin and subcutaneous tissue disorders) | 75 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 108 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 44 | 24
Rash (Skin and subcutaneous tissue disorders) | 109 | 39
Skin discolouration (Skin and subcutaneous tissue disorders) | 94 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 37 | 5
Hypertension (Vascular disorders) | 125 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.